# THE UNIVERSITY OF TEXAS M. D. ANDERSON CANCER CENTER

#### **DIVISION OF MEDICINE**

FLUDARABINE, MITOXANTRONE, AND DEXAMETHASONE (FND) PLUS CHIMERIC ANTI-CD20 MONOCLONAL ANTIBODY (RITUXIMAB) FOR STAGE IV INDOLENT LYMPHOMA

| | ABSTRACT |
|---|---|
| 1.0 | OBJECTIVES |
| 2.0 | INTRODUCTION |
| 3.0 | BACKGROUND DRUG INFORMATION |
| 4.0 | PATIENT ELIGIBILITY |
| 5.0 | TREATMENT PLAN |
| 6.0 | PRETREATMENT EVALUATION |
| 7.0 | EVALUATION DURING STUDY |
| 8.0 | CRITERIA FOR RESPONSE AND TOXICITY |
| 9.0 | CRITERIA FOR REMOVAL FROM STUDY |
| 10.0 | STATISTICAL CONSIDERATIONS |
| 11.0 | DATA AND PROTOCOL MANAGEMENT |
| 12.0 | REPORTING REQUIREMENTS |
| 13.0 | REFERENCES |
| | APPENDICES Appendix A: Activity Flow Chart Appendix B: Management Strategy for Follicular Lymphoma Patients Who Do Not Have bcl-2 mbr or mcr Gene Rearrangement ("Germline" Patients) Appendix C: Performance Status Criteria Appendix D: Adult Toxicity Criteria Appendix E: Directions for Preparing Rituximab Administrations Appendix F: Additional Safety Guidelines for Use of Interferon Appendix G: Guidelines for Reporting ADRs to the IRB Appendix H: Adverse Events Reporting (MEDWATCH Form) Informed Consent |
| | HIOTHICA COMMENT |

Peter McLaughlin, M.D.

STUDY CHAIRMAN:

## **COLLABORATORS:**

11

Fernando Cabanillas, M.D.

M. Alma Rodriguez, M.D.

Andreas H. Sarris, M.D., Ph.D.

Ming-Sheng Lee, M.D.

Shirley Riggs, M.D.

Terry Smith, A.S.

Fredrick B. Hagemeister, M.D.

Jorge Romaguera, M.D.

Anas Younes, M.D.

Donna Weber, M.D.

Nam H. Dang, M.D., Ph.D.

## **COLLABORATORS:**

| Fernando Cabanillas, M.D. | Fredrick B. Hagemeister, M.D. |
|--------------------------------|-------------------------------|
| M. Alma Rodriguez, M.D. | Jorge E. Romaguera, M.D. |
| Andreas H. Sarris, M.D., Ph.D. | Anas Younes, M.D. |
| Ming-Sheng Lee, M.D. | Donna Weber, M.D. |
| Nam Dang, M.D., Ph.D. | Terry Smith, B.S. |

The University of Texas M.D. Anderson Cancer Center Department of Lymphoma/Myeloma 1515 Holcombe Blvd., Box 429 Houston, TX 77030

#### PROTOCOL ABSTRACT

PROTOCOL: (Abbreviated title) (2 lines/75 characters per line) (USE 12 PT ONLY)

Fludarabine, Mitoxantrone, and Dexamethasone (FND) Plus Anti-CD20 Monoclonal Antibody (rituximab) for Stage IV Indolent Lymphoma

STUDY CHAIRMAN

Peter McLaughlin, MD

#### **OBJECTIVES:**

- 1. To compare molecular response rates with the FND regimen followed by rituximab (chimeric anti-CD20 antibody) and interferon versus FND plus rituximab concurrently, followed by interferon, for patients with stage IV indolent lymphoma.
- 2. To compare the toxicity of these two regimens, including their effects on B- and T- cell subsets, immunoglobulins, and patterns of infections.
- 3. To compare failure-free and overall survival rates with these two regimens.
- 4. To identify and treat with a separate strategy those follicular lymphoma patients without bcl-2 mbr or mcr gene rearrangement ("germline" patients) because of their adverse outcome with FND alone in our prior experience.

#### RATIONALE: (Be as concise as possible)

For all stage IV indolent lymphomas (with one exception; see Appendix B), the FND regimen appears to be comparable to the more intensive ATT regimen, in terms of remission rates, failure-free survival, and even molecular remission rates. The anti-CD20 monoclonal antibody rituximab is a promising agent with modest toxicities, none of which should overlap with the toxicities of FND. Hence, we propose to combine FND + rituximab, either concurrently or with rituximab as post-FND adjuvant therapy.

#### ELIGIBILITY: (List Major Criteria)

- Previously untreated stage IV indolent B-cell lymphoma [Amendment May 2001: eligibility restricted to <u>follicular</u> lymphoma]
- Age <76

#### TREATMENT PLAN:

| Γ | I. FND | | | | |
|---|---|---|---|---|---|
| ١ | Fludarabine | $25 \mathrm{mg/m^2}$ | IV | qd x 3 d1-3 | (d2-4 in conjunction with IDEC) |
| l | Novantrone | $10\mathrm{mg/m^2}$ | IV | day 1 only | (day 2 only in conjunction with IDEC) |
| ı | Decadron | 20 mg | IV | qd x 5 | d1-5 |

II. Rituximab 375 mg/m² per dose

Dosing and schedule integrated with FND (see Section 5.3) or after FND (see section 5.2.3)

III. Interferon alfa-2b maintenance  $3 \times 10^6$  U/m²/d x 14 days 1-14 of each 28 day maintenance cycle for 12 cycles, with decadron 8 mg qd x 3, days 1-3. (see Section 5.7.3 for integration of IFN cycles with rituximab)

#### STATISTICAL CONSIDERATIONS:

The average yearly accrual rate for the current stage IV trial has been 33 patients per year. About 75% of patients can be expected to have a positive PCR. It will take 64 PCR positive patients in each arm to detect a difference of 25% in the twelve month molecular CR rate, assuming that the higher response rate was 85%. This assumes a two-sided alpha level of 0.05 and a power of 0.90.

Allowing for some inevaluable cases, approximately 210 patients will be accrued, which will probably take a little over 5 years.

PATIENT EVALUATION: (Pretreatment and Interim Testing)

| TATILITY LV | ILIOTITIO | 1. (1 1 C L C C C C C C C C C C C C C C C C | | CIMIT TESTING) | TIX /TIDA / | |
|---|---|---|---|---|---|---|
| | | | EVERY | EVERY | EVERY | |
| 1 | PRE | | 2 | 3 | 6 | POST- |
| l | STUDY | WEEKLY | <b>COURSES</b> | COURSES | <b>MONTHS</b> | <b>THERAPY</b> |
| H&P | X | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | X | 3-7-2-3-3-3-3-3-3-3-3-3-3-3-3-3-3-3-3-3- | · | q 3-6 mo |
| PS | X | | | | | |
| CBC | X | X | | | | q 3-6 mo |
| U/A | X | | | | | , |
| CXR | X | | | | | q 3-6 mo <sup>‡</sup><br>q 3-6 mo |
| SMA 12, K, Mg* | X | | X | | | q 3-6 mo |
| B2M | X | | | X | | q 3-6 mo |
| BX/FNA* | X | | | | | , |
| BM BX | X | | | X | | q 6 mo <sup>‡</sup><br>q 6 mo <sup>‡</sup> |
| LAG, CTs | X | | | X | | q 6 mo‡ |
| PB markers, Ig's | X | | | X*** | | |
| PB PCR | X | | | | X** | |
| BM PCR | X | | | | X** | |
| ECHO or MUGA | X | | | | | |

- \* K, Mg, etc as indicated, mainly for pts on ATT (see App. B)
- \* when accessible; for phenotype, gene rearrangement
- \*\* PCR for bcl-2 q 6 mo yr 1-3, q 12 mo thereafter. Contingency for PCR monitoring at 9 and/or 15 months for selected patients (see 7.2).

\*\*\* PB markers, Ig's: until recovery to normal

‡ Restaging off therapy (see section 7.7): at least q 6 mo until relapse or through year 5; then at least yearly

MISCELLANEOUS INFORMATION: (Include any other information that you feel is pertinent to the study) (Three lines not to exceed 75 characters per line)

- PCP prophylasix: TMP/SMX, 2 DS tabs PO twice weekly (q Sat & Sun). For allergy, see section 5.4.3.2
- If PCP pneumonia occurs, subsequent chemotherapy cycles will be given without dexamethasone.

| ESTIMATED ACCRUAL: |
|---|
| It is estimated that accrual will be2 participants per month. |
| SITE OF STUDY: (please circle the appropriate answer) |
| This protocol is performed on an:INPATIENT BOTH basis |
| LENGTH OF STAY: (What is the length and frequency of hospitalization) |
| RETURN VISITS: (How often must participants come to MDACC) |
| TELECTICAL VICTOR CITICAL PLANTS CONTROL CONTR |
| HOME CARE: (specify what (if any) treatment may be given at home) |
| WHERE THE STUDY WILL BE CONDUCTED: |
| A) ONLY AT MDACC B) MDACC + COMMUNITY PROGRAMS C) INDEPENDENT (CCOP, NETWORK) MULTICENTER ARRANGEMENTS |
| NAME OF SPONSOR/FUNDING SOURCE: |
| COMPETING PROTOCOLS: (Protocol number(s)) |
| NONE |
| NAME OF RESEARCH NURSE/DATA MANAGER RESPONSIBLE FOR PROTOCOL: |

#### SUBMIT PROTOCOL TO CLINICAL RESEARCH CENTER REVIEW COMMITTEE:

YES D NO D

IF YOUR PROTOCOL HAS A DIAGNOSTIC STEP REQUIRING INFORMED CONSENT AND REGISTRATION ON THE PROTOCOL (E.G., A BLOOD TEST OR BIOPSY) THAT WILL DETERMINE WHETHER OR NOT THE PATIENT WILL SUBSEQUENTLY RECEIVED OR NOT RECEIVED EXPERIMENTAL THERAPY. PLEASE CHECK THE APPROPRIATE BOX(ES) SO THAT THE APPROPRIATE FIELDS MAY BE ESTABLISHED IN PDMS:

BLOOD TEST: YES NO BIOPSY: YES NO OTHER: YES NO

The University of Texas

M. D. Anderson Cancer Center OFFICE OF PROTOCOL RESEARCH

PROTOCOL APPROVED

# THE UNIVERSITY OF TEXAS M. D. ANDERSON CANCER CENTER



#### **DIVISION OF MEDICINE**

FLUDARABINE, MITOXANTRONE, AND DEXAMETHASONE (FND) PLUS CHIMERIC ANTI-CD20 MONOCLONAL ANTIBODY (RITUXIMAB) FOR STAGE IV INDOLENT LYMPHOMA

#### **ABSTRACT**

- 1.0 OBJECTIVES
- 2.0 INTRODUCTION
- 3.0 BACKGROUND DRUG INFORMATION
- 4.0 PATIENT ELIGIBILITY
- 5.0 TREATMENT PLAN
- 6.0 PRETREATMENT EVALUATION
- 7.0 EVALUATION DURING STUDY
- 8.0 CRITERIA FOR RESPONSE AND TOXICITY
- 9.0 CRITERIA FOR REMOVAL FROM STUDY
- 10.0 STATISTICAL CONSIDERATIONS
- 11.0 DATA AND PROTOCOL MANAGEMENT
- 12.0 REPORTING REQUIREMENTS
- 13.0 REFERENCES

#### **APPENDICES**

Appendix A: Activity Flow Chart

Appendix B: Management Strategy for Follicular Lymphoma Patients Who Do Not

Have bcl-2 mbr or mcr Gene Rearrangement ("Germline" Patients)

Appendix C: Performance Status Criteria

Appendix D: Adult Toxicity Criteria

Appendix E: Directions for Preparing Rituximab Administrations Appendix F: Additional Safety Guidelines for Use of Interferon

Appendix G: Guidelines for Reporting ADRs to the IRB

Appendix H: Adverse Events Reporting (MEDWATCH Form)

Informed Consent

STUDY CHAIRMAN:

Peter McLaughlin, M.D.

#### 1.0 OBJECTIVES

- 1.1 To compare molecular response rates with the FND regimen followed by rituximab (chimeric anti-CD20 antibody) and interferon versus FND plus rituximab concurrently, followed by interferon, for patients with stage IV indolent lymphoma.
- 1.2 To compare the toxicity of these two regimens, including their effects on B- and T-cell subsets, immunoglobulins, and patterns of infections.
- 1.3 To compare failure-free and overall survival rates with these two regimens.
- 1.4 To identify and treat with a separate strategy those follicular lymphoma patients without bcl-2 mbr or mcr gene rearrangement ("germline" patients) because or their adverse outcome with FND alone in our prior experience.

#### 2.0 BACKGROUND

#### 2.1 The Disease

The indolent lymphomas are characterized by a slow pace, typically by responsiveness to at least the initial therapy, but by inevitable relapse following standard therapy.

The histologic categories that comprise the majority of cases of indolent lymphoma are small lymphocytic lymphoma (SL), follicular small cleaved (FSC), and follicular mixed (FM) lymphoma as defined in the Working Formulation<sup>1</sup>. However, it is notable that the recent Revised European American Lymphoma (REAL) scheme has: (a) created a scheme that more precisely categorizes several subsets of SL, including mantle cell lymphoma (MCL) which is considered not indolent; (b) challenged the concept that follicular large cell lymphoma (FLC) is intermediate grade and classifies FLC (follicle center lymphoma, follicular, grade III) along with the other follicular lymphomas.

Concerning subsets that have previously been categorized as SL: (a) we currently have a separate treatment strategy for MCL; (b) MALT lymphomas, when they present with localized disease, have a separate appropriate treatment strategy; but (c) when the marginal cell lymphomas present with disseminated disease, they are just as relentless as other advanced stage indolent lymphomas<sup>3</sup> and therefore deserve, in our opinion, the same treatment strategy as other advanced stage indolent lymphomas.

Concerning FLC, inter-institutional and inter-pathologist differences in classification are well known for subclassification of follicular lymphomas<sup>4</sup>. At MDACC, the distinction between follicular large non-cleaved versus cleaved lymphoma has been emphasized in recent years<sup>5</sup>, the latter being considered indolent and thus eligible for this protocol, while the former is considered aggressive and such cases are triaged to other protocols. It is acknowledged that the distinction among precise cell types among the follicular lymphomas is at times arbitrary. Pertinent to therapy considerations (see below), FLC is unique among the intermediate grade lymphomas in that responsiveness to fludarabine is typically good<sup>6</sup>.

An important hallmark of the follicular lymphomas is the t(14;18) translocation which results in bcl-2 gene rearrangement in the majority of cases. Among other things, this breakpoint provides a marker that can be followed by PCR (see below). There is beginning to be evidence that the specific breakpoint site (mbr; mcr) may be prognostically important, and the "germline" (i.e., not mbr or mcr rearranged) cases may do poorly with FND chemotherapy. Accordingly, in this protocol such patients are assigned to a separate treatment strategy

2.2 Chemotherapy Approaches

Using therapy based on alkylating agents such as cyclophosphamide and chlorambucil, depressingly little has changed in survival outcomes in the past 30 years<sup>8</sup>. In the intermediate grade lymphomas, the impact of doxorubicin is compelling<sup>9</sup>; but the impact of the addition of doxorubicin in indolent lymphoma is arguable <sup>9,10</sup>. To date, the impact of interferon (IFN) appears mainly on duration of remission rather than on survival<sup>11</sup>. The purine nucleoside analogs, especially fludarabine, are a new class of drugs that have appeared very promising in indolent lymphoma and chronic lymphocytic leukemia<sup>6</sup>. Fludarabine has been used extensively in relapsed indolent lymphoma, both singly and in combination regimens<sup>6</sup>. At MDACC, the FND regimen has been used successfully in front-line therapy, with early results showing it to be comparable to the more intensive "ATT" regimen<sup>12,13</sup>. One subset of follicular lymphoma for whom FND may be inferior to ATT are those with "germline" status for bcl-2<sup>7</sup>.

#### 2.3 PCR for bcl-2

The initial description of the utility of PCR for bcl-2 in detecting the subclinical presence of rearranged cells was here at MDACC. Since then, the role of this assay as a surrogate endpoint and marker of treatment success has generated worldwide interest<sup>15-17</sup>.

The attainment of PCR-negativity with any therapy approach except bone marrow transplantation has been difficult<sup>18,19</sup>. In recent years, reversion to PCR-negativity has been accomplished with our "ATT" regimen<sup>13</sup>. Thus, it is possible to explore whether attaining PCR-negativity is a desirable goal that correlates with more durable remission, as has been observed with bone marrow transplantation and *ex vivo* purging<sup>15,19</sup>. Our preliminary results indicate that PCR-negativity does indeed correlate with longer remission following conventional dose chemotherapy<sup>20</sup>.

Our recent experience (DM 92-103) with FND has shown that this regimen, too, can induce PCR-negativity<sup>12</sup>. The current protocol is a logical extension of that experience.

#### 2.4 Anti-CD20 Monoclonal Antibody Therapy (rituximab)

Monoclonal antibodies are of tremendous theoretical appeal as therapeutic agents. Our understanding of the expression of surface antigens in B-cell malignancies has led to numerous trials of monoclonal antibodies in B-cell malignacies<sup>21</sup>. Stumbling blocks have been encountered, including the immunogenicity of rodent monoclonal antibodies and the myelosuppressive effects of radioimmunoconjugates.

A chimeric anti-CD20 antibody, rituximab, has emerged as a promising single agent. Since it is predominantly a human protein, host immune responses against the agent have been infrequent. Since it is not conjugated to a toxin or isotope, its spectrum of toxicity is relatively modest. And, most importantly, as a single agent

is has been shown to have promising activity in patients with relapsed B-cell lymphoma<sup>22,23</sup>.

Rituximab has been used in conjunction with standard CHOP chemotherapy, with promising early results<sup>24</sup>. Other combination trials, including the current protocol, are planned.

The most extensive experience with rituximab, as a single agent, has utilized a schedule of weekly dosing for four weeks. Its relative lack of immunogenicity suggests that re-treatment or longer-term treatment schedules are feasible. This issue is to be explored in one arm of the current trial.

The experience with rituximab in conjunction with CHOP chemotherapy utilized a total of six doses of the antibody, integrated into the chemotherapy cycles in a fashion similar to the other proposed arm of our current protocol. This integration of rituximab with chemotherapy has already been shown feasible and effective with CHOP. The current protocol will be the initial experience of the integration of rituximab with the FND regimen.

Rituximab appears to be capable of effecting reversion of PCR for bcl-2 in the peripheral blood and bone marrow from positive to negative. Using the antibody alone, the peripheral blood became PCR-negative in 68% and the bone marrow in 50% <sup>23</sup>. In conjunction with CHOP, the peripheral blood became PCR-negative in almost 80% <sup>24</sup>. Since CHOP alone appears to result in PCR-negativity only infrequently, the expectation of higher rates of PCR negativity, coupled with in vitro evidence of synergism between rituximab and some chemotherapeutic agents <sup>25</sup>, warrants further experience with concurrent antibody plus chemotherapy.

Given the potential of rituximab to produce, as a single agent, PCR negativity in the blood and marrow <sup>26</sup>, and since some chemotherapy-treated patients do <u>not</u> achieve PCR negativity, the adjuvant use of the antibody may result in higher molecular remission rates (although at a later time point than 12 months). This potential for eradication of minimal residual disease, and extrapolation from our previous favorable experience with adjuvant interferon, provide the rationale for the adjuvant antibody strategy.

As previously discussed, a small subset of patients with follicular lymphoma are germline for bcl-2, and our experience suggests that these patients may be prognostically unfavorable, in that an intensive regimen such as ATT appears necessary for best results. For these patients, we propose integration of rituximab with ATT.

#### 3.0 BACKGROUND DRUG INFORMATION

- 3.1 For fludarabine, mitoxantrone, dexamethasone, interferon alfa-2b (Intron A), and the agents in the CHOD-Bleo/ESHAP/NOPP program, data available on request (713-792-2860).
- 3.2 Rituximab chimeric anti-CD20 antibody.

3.2.1 Investigational Drug Nomenclature

• IDEC Pharmaceuticals code designation: IDEC-C2B8 (IDEC-102)

• Generic name: Rituximab

CAS Registry number: 174722-31-7

• IND number: BB-IND 4904

3.2.2 Origin of the IDEC-C2B8 cell line.

The chimeric mouse/human anti-CD20 monoclonal antibody, rituximab (IDEC-C2B8 [IDEC-102]), is a human gamma 1 kappa antibody with mouse variable regions isolated from a murine anti-CD20 monoclonal antibody (2B8). This chimeric antibody, which is secreted by the Chinese hamster ovary (CHO) transfectoma clone 8-8F12-5E5-50C9, binds with high affinity to CD20-positive cells, performs human effector functions in in vitro assays, and specifically depletes B cells in vivo. The CHO transfectoma was produced by inserting DNA coding for the chimeric immunoglobulin chains into the CHO cell line DG44 by electroporation, and selecting for a clone resistant to G418 (Genetecin) that secreted chimeric immunoglobulin (Clone 8-8F12). Subsequently, the immunoglobulin production was enhanced through selection of a clone resistant to 5 nM methotrexate (MTX) (clone 8-8F12-5E5); Phase I and Phase II material was produced using this clone. Immunoglobulin production was further enhanced through selection of a clone resistant to 50nM MTX (clone 8-8F12-5E5-50C9). Material produced from this clone has been used in a Phase II combination study with CHOP.

3.2.2.1 Development Code: IDEC-C2B8 (IDEC-102)

3.2.2.2 Other Designations: Mouse/human chimeric monoclonal antibody for CD20 antigen; anti-CD20 antibody, chimeric pan-B.

#### 3.2.3 Clinical Formulation

Clinical supplies for this study will be manufactured by either IDEC Pharmaceuticals in San Diego, CA or Genentech Incorporated in South San Francisco, CA.

Rituximab from either source will be provided to the clinical sites packaged in single use 10 mL (100 mg) and 50mL (500 mg) Type I glass vials at a concentration of 10 mg of protein per mL. The product is formulated in 7.35 mg/mL sodium citrate buffer, containing 7 mg/mL polysorbate 80, 9.0 mg/mL sodium chloride and Sterile Water for Injection. The pH is adjusted to 6.5.

Rituximab may be produced by the mammalian (Chinese Hamster Ovary) cell suspension culture in a nutrient medium containing 100 mg/mL of the antibiotic gentamicin. The antibiotic is not detectable in the final product.

3.2.4 Storage

Rituximab for clinical use should be stored in a secure refrigerator at 2-8° C.

3.2.5 Reconstitution and Dilution of rituximab
Using a sterile syringe and a 21 gauge or larger needle, transfer the
necessary amount of rituximab from the vial into a partially filled IV pack
containing sterile, pyrogen-free 0.9% Sodium Chloride, USP (saline
solution). The final concentration of Rituximab should be approximately 1
mg/mL. Mix by inverting the bag gently.

For lots 0122-0125 the final preparation should be administered through a 0.22 micron low-protein binding in line filter, such as IMED 9216, into the outflow port of the bag containing the infusion solution. For other lots this will not be required.

Caution should be taken during the preparation of the drug. (See Appendix I). Parenteral drug products should be inspected visually for particulate matter prior to administration, Preparations of rituximab containing visible particles should note be used. As with all parenteral drug products, aseptic procedures should be used during the preparation and administration of rituximab.

NOTE: DO NOT USE A VACUUM APPARATUS to transfer rituximab from the syringe to the infusion pack. DO NOT USE evacuated glass container which require vented administration sets, because this causes foaming when air bubbles pass through the solution.

# 3.2.6 Product Administration

In calculating body surface area, actual height and weight should be used, that is, there will be no downward adjustment to "ideal" weight. <u>Dosage calculations for all treatments will be calculated using the patient's body surface area as determined during the screening evaluation.</u> The dose level of rituximab will not be adjusted.

#### 3.2.7 Pre-Clinical Experience

Rituximab (IDEC-102) is a chimeric IgG1 kappa monoclonal antibody, with mouse variable and human constant regions, that recognizes the CD20 antigen expressed on normal B cells and most malignant B-cell lymphomas<sup>1</sup>. The antigen, important in cell cycle initiation and differentiation, is expressed strongly in over 90% of B-cell lymphomas. Rituximab shows specificity for the CD20 antigen and binds with an apparent affinity of  $5.2 \times 10^{-9}$ M.

In vitro mechanism of action studies have demonstrated that this antibody binds human complement and lyses lymphoid B cell lines. It has significant activity in assays for antibody-dependent cellular cytotoxicity (ADCC). High dose safety studies in cynomolgus monkeys revealed a decrease in platelet levels between 7 and 33% at the two higher doses on day 1 with recovery between days 7 and 14. A reduction in white blood cells between 13 and 31% was seen in 5 of 6 monkeys studied with recovery beginning by day 8. In 4 of 6 monkeys at 12 to 34% decrease in segmented neutrophils was observed; recovery occurred by day 14 in one animal. Hematologic changes were not dose-dependent. In this study and during other rituximab testing in cynomolgus monkeys, vomiting

was noted in a minority of monkeys. Dose levels of 20 mg/kg weekly for up to eight weeks showed no significant adverse reactions, toxicological events or any abnormal histopathology. The biologic effect of four weekly doses of rituximab in cynomolgus monkeys resulted in B-cell depletion in peripheral blood (PB), lymph nodes (LN) and bone marrow (BM). Three weeks after 4 weekly doses there was a >75% decrease of B cells in the bone marrow. Recovery of the B cells in the peripheral blood (to >75% of baseline) usually occurred within 60 days following the last dose.

#### 3.2.8 Clinical Experience

Previous clinical trials have shown that outpatient therapy with rituximab, completed within 22 days, is safe and effective in the treatment of patients with relapsed low-grade/follicular non-Hodgkin's lymphoma.

#### Phase I/II Trials

Two previous Phase I/II dose-escalation studies of rituximab were conducted (IDEC Protocols 102-01 and 102-02) in patients with relapsed or recurrent non-Hodgkin's lymphoma [Maloney, 1994#1537;[3]. Fifteen patients were enrolled in a single-dose study (IDEC 102-01), (10 to 500 mg/m<sup>2</sup> of rituximab) and 47 patients in a multiple-dose study (IDEC 102-02) (125, 250, or 375 mg/m2 once weekly times four). Clinical activity was noted in seven of 15 patients in the single-dose trial with two partial responses lasting 8.1 and 8.5 months, and five minor responses lasting between 0.9 and 6 months. In the multiple-dose study, three complete responses and 14 partial responses were noted in 34 evaluable patients  $(375 \text{ mg/m}^2 \text{ rituximab})$  with a median response duration of 8.6 months. Median time to progression (TTP) in responders was 10.2 months; TTP exceeded 20 months in five patients, two of whom have ongoing responses of 30+ months. No correlation between pharmacokinetic parameters clinical response was apparent in the single-dose study; however, a positive correlation was observed between clinical response and antibody serum levels prior to the second infusion in the multipledose study.

Overall, adverse experience were mostly Grades 1 and 2 and consisted primarily of infusion-related events (fever, asthenia, chills, headache, and less commonly, bronchospasm, hypotention and agioedema[subjective sensation of tongue and throat swelling). Hematologic toxicity was usually mild and reversible. In both trials, a rapid an selective depletion of circulating B-cells was observed following treatment. In the Phase I/II study, mean serum immunoglobulin levels remained stable, although some patients experienced transient reductions of IgOs. In both studies, it was concluded that intravenous infusions of rituximab appeared safe and well tolerated and demonstrated significant activity in patients with relapsed B-cell lymphoma.

#### Phase III Open-Label Trial

A Phase III multicenter trial completed patient entry in March 1996 with a total enrollment of 166 patients [4]. Treatment consisted of weekly x four infusions at 375 mg/m². Analysis revealed that adverse events (AE) were primarily related to first infusion and consisted of fever, chills, nausea, and headache. There was a marked reduction in the incidence of AEs in

subsequent infusions. Overall, 6% of all events (72 of 1163) observed during study treatment and follow-up were Grade 3 and 4, and of those, 3% (39 of 1163) were related to study treatment. There were no incidences of human antichimeric antibody (HACA) during this trial. (The overall incidence of HACA in over 300 patients participating in all rituximab trials has been <1% and HACA was not clinically significant in those in whom it occurred).

Ninety-one percent of patients (151 of 166) were evaluable for efficacy and achieved an overall response rate of 50% with 6% CR and 44% of PR. The onset of response was as early as even weeks and responses were seen in patients with bulky and extranodal disease. CT scans of responders were reviewed and confirmed (blinded audit) by an independent panel of lymphoma experts following established response criteria. Median time to progression for responders had not been reached with 9+ months median follow-up.

#### 4.0 ELIGIBILITY

- 4.1 Previously untreated patients, younger than 76 years old, with stage IV follicular lymphoma (including follicular large cleaved cell) or small lymphocytic lymphoma. [Amendment May 2001: Eligibility for last 25-30 patients restricted to follicular lymphoma (see section 10.2)]
  - 4.1.1 Patients with chronic lymphocytic leukemia (absolute lymphocyte count >5000 μL) are excluded.
  - 4.1.2 Patients with divergent histologies (intermediate grade in one site and low grade in another) will not be eligible.
  - 4.1.3 It is known that there can be a continuum of histologies, spanning elements of indolent and aggressive. While patients with truly divergent histologies are specifically excluded (see 4.1.2), other variants can be eligible, as follows:
    - F + DSC\* eligible.
    - F + DM\* eligible.
    - Sclerosing SCCL or mixed cell eligible (even if follicular architecture not definite)
    - Follicular large noncleaved cell the distinction between this entity and follicular large cleaved can be arbitrary and is of debatable significance. But it has been our practice to treat follicular large noncleaved as an intermediate grade lymphoma. Hence, if eligible, such patients should be treated on the appropriate intermediate grade protocol. However, both FND and rituximab have established efficacy in FLCL (without regard to cleaved or not), so if a patient is not eligible for an intermediate grade protocol (e.g., because of SCCL in the marrow), then registration on this trial is permitted.
    - FSC or FM with areas of FLC eligible.
    - FSC or FM with areas of DLC <u>not</u> eligible unless reviewed with P.I. and an addendum on the pathology report is issued stating that the disease is best categorized as an indolent lymphoma.

- \*- in F & D cases, <u>any</u> extent of follicular architecture is traditionally accepted, but in cases that are > 75% diffuse, please review with P.I. and Pathology as for 4.1.3 (f) above.
- 4.2 Patients must sign an informed consent indicating that they are aware of the invitational nature of the study, in keeping with the policies of the hospital.
- 4.3 Ineligible patients are:
  - 4.3.1 Patients who are unable or unlikely to be able to adhere to the treatment plan or to return to Houston for follow-up visits because of geographical, economic, emotional, or social considerations are not eligible for this study.
  - 4.3.2 Patients with an absolute peripheral granulocyte count of < 1,000 and platelet count < 100,000 unless due to marrow infiltration or hypersplenism.
  - 4.3.3 Patients with hepatic dysfunction, defined as bilirubin of > 1.5 mg%, unless the alteration is due to lymphoma.
  - 4.3.4 Patients with a serum creatinine level >1.5 mg% unless the alteration is due to lymphoma.
  - 4.3.5 Patients with HIV infection should not be registered on this protocol.
  - 4.3.6 Pts with an antecedent malignancy whose prognosis is poor (< 90% probability of surviving for 5 yrs).
  - 4.3.7 All patients should have a cardiac ejection fraction of ≥ 50% by echocardiography or MUGA. If a patient without cardiac symptoms has an aberrant low LVEF (< 50%), please consult cardiology and discuss with P.I.
  - 4.3.8 Patients who will not accept transfusions of blood products or supportive care measures such as antibiotics are not eligible for this study.
  - 4.3.9 Female patients must not be pregnant or lactating, and men and women of reproductive potential must follow accepted birth control methods.
- 4.4 Additional safety guidelines for use of interferon (see Appendix F): These considerations are not exclusions to eligibility since:
  - (1) Some abnormalities might change before IFN maintenance, e.g., organ dysfunction related to disease might likely improve with treatment; or
  - (2) some guidelines, e.g., a history of depression, might mitigate against IFN but would <u>not</u> exclude the patient's being treated on protocol with all the other elements of the program.

Please discuss any concerns about IFN with the P.I.

#### 5.0 TREATMENT PLAN

5.1. All patients must be registered with Data Management at 792-2926. They will be interviewed first by the Research Nurse before registration.

5.1.1 Follicular lymphoma patients who are known not to have bcl-2 gene rearrangement will <u>not</u> be randomized -- they will proceed directly to therapy with the ATT regimen (see Appendix B).

If there is no threatening disease and the clinician judges that it is safe to wait for the bcl-2 data, the initiation of therapy may be delayed (This is encouraged.)

However, if therapy is needed, it will not be delayed just for the bcl-2 report. If bcl-2 status is not known or pending, patients <u>will</u> be randomized. If, after therapy with FND begins, a patient is found to be germline for bcl-2, the patient will be crossed over to ATT (see strategy outline in Appendix B).

- 5.1.2 Randomization will be stratified for: tumor mass size < 5 cm vs. ≥ 5 cm; age < 60; FLC histology; SL histology; and suitability for the watch-and-wait policy followed at other institutions.
- 5.2 <u>ARM 1 (delayed anti-CD20 arm)</u> will consist of consecutive courses of Fludarabine/Mitoxantrone/Dexamethasone (FND), followed by rituximab.

| <u>Agent</u> | <u>Dose</u> | <u>Days</u> | <u>Route</u> | <u>Time</u> | Total Dose |
|---|---|---|---|---|---|
| Fludarabine | 25 mg/m <sup>2</sup> | 1-3 | IV | 15 min | 75 mg/m <sup>2</sup> |
| Mitoxantrone | 10 mg/m <sup>2</sup> | 1 | IV | 15 min | 10 mg/m <sup>2</sup> |
| Decadron | 20 mg | 1-5 | IV or PO | 15 min | 100 mg |

5.2.1 Duration of therapy and intervals between courses:

a) The courses should be repeated every 28 days according to recovery from

myelosuppression.

- b) The total length of treatment will be 8 courses unless cumulative myelosuppression is encountered, in which case the treatment will be finished after 6 courses. Cumulative myelosuppression is defined as recovery of granulocytes to ≥ 1,000 or platelets to >100,000 requiring more than 6 weeks.
- 5.2.2 Patients older than 60 years will receive full doses of chemotherapy. Anyone experiencing delayed recovery of granulocyte counts (>35 days) or neutropenic fever will be candidates for G-CSF (Neupogen), with the chemotherapy doses adjusted down one dose level. The G-CSF dose will consist of 300 mcg total dose daily, subcutaneously. The dose can be increased to 480 mcg daily at the clinician's discretion.
- 5.2.3 Rituximab Adjuvant Therapy Starting at 12 months, after collection of the 12-month PCR samples (Sec 7.2), rituximab will be given monthly for 6 doses total.

The dose will be 375 mg/m² IV. Interferon maintenance will usually have commenced about 3-4 months before the rituximab doses start. When IFN and rituximab doses are given in the same month, the rituximab dose will be given first, with decadron permitted (but not mandatory) and the IFN will begin on day 2 of each cycle, or may be delayed for 1-2 days if needed (see 5.7.3).

When rituximab is given by itself (without IFN), decadron 8 mg IV or PO as a pre-medication is permitted but not mandatory (and see also 5.4).

5.3 <u>ARM 2</u> (concurrent anti-CD20 arm) will consist of FND in conjunction with rituximab. Rituximab will be given on days 1 and 8 of course 1, then on day 1 only of courses 2-5, as outlined below:

#### - course 1:

rituximab 375 mg/m² d.1 & 8 IV (see section 5.4 for details of administration) fludarabine 25 mg/m² d. 2-4 IV mitoxantrone 10 mg/m² d.2 IV dexamethasone 20 mg d. 1-5 IV or PO (note dexamethasone starts a day earlier than in the usual FND schedule, so that the first dose of rituximab is given in conjunction with steroid)

#### - courses 2-5:

rituximab 375 mg/m $^2$  d.1 IV (see section 5.4 for details of administration) fludarabine 25 mg/m $^2$  d. 2-4 IV mitoxantrone 10 mg/m $^2$  d.2 IV dexamethasone 20 mg d. 1-5 IV or PO (note dexamethasone starts a day earlier than in the usual FND schedule, so that the first dose of rituximab is given in conjunction with steroid)

#### - courses 6 - 8:

same as for arm 1 (i.e., FND without concurrent rituximab) -- see Section 5.2, especially 5.2.1 and 5.2.2 concerning interval (q28 d), guidelines for use of G-CSF (applicable for <u>all</u> courses), and guidelines for omitting courses 7 & 8 if there is cumulative myelosuppression

#### 5.4 Details Pertaining to Rituximab Administration

#### 5.4.1 Rituximab Dose

All patients enrolled into the study will receive fixed doses of rituximab at 375 mg/m². In calculating body surface area, actual height and weight should be used, that is, there will be no downward adjustment to "ideal" weight. Dosage for all treatments will be calculated using the patient's body surface area as determined during the baseline evaluation. The dose level of rituximab will <u>not</u> be adjusted thereafter.

#### 5.4.2 Method of Administration

# CAUTION: DO NOT ADMINISTER AS AN INTRAVENOUS PUSH OR BOLUS.

Rituximab infusions will be administered to patients in an outpatient clinic setting. To decrease the incidence of infusion-related adverse events, oral premedication (650 mg of acetaminophen and 25-50 mg diphenhydramine hydrochloride) may be administered prior to starting

each infusion of rituximab. Decadron 8 mg IV or PO is also permitted. A peripheral or central intravenous (IV) line will be established. During the rituximab infusion, the patient's vital signs (blood pressure, pulse, respiration, temperature) should be monitored every 15 minutes x 4 or until stable and then hourly until the infusion is discontinued.

Available at the bedside prior to rituximab administration will be:

- (a) epinephrine for subcutaneous injection;
- (b) diphenhydramine hydrochloride for intravenous injection; and
- (c) resuscitation equipment for the emergency management of anaphylactoid reactions.

The initial dose rate at the time of the first rituximab infusion should be 50 mg/hr for the first hour. If no toxicity is seen, the dose rate may be escalated gradually (50 mg/hr increments at 30-minute intervals) to a maximum of 400 mg/hr. If the first dose of rituximab is well tolerated, the starting flow rate for the administration of subsequent doses will be 100 mg/hour then increased gradually (100 mg/hr increments at 30-minute intervals) not to exceed 400 mg/hr.

Since transient hypotention has been reported during rituximab infusions, consideration should be given to withholding anti-hypertensive medications the day of the rituximab infusion. Patients may experience transient fever and rigors with rituximab. When these side effects are noted, the antibody infusion should be temporarily slowed or discontinued, the patient should be observed, and the severity of the side effects should be evaluated. The patient should be treated according to the best available local practices and procedures. Following observation, when the patient's symptoms improve, the infusion should be continued, initially at 1/2 the previous rate and gradually escalated to a maximum rate of 300 mg/hour (see table below). Following the antibody infusion, the IV line should be kept open for medications, as needed. If there are no complications, the IV line may be discontinued after one hour of observation. If complications occur during the rituximab infusion, the patient should be observed for two hours after the completion of the infusion.

In patients with detectable circulating lymphoma cells, it is strongly advised that the initial rate of infusion be reduced to 25 mg/hr. Patients with detectable circulating cells may experience more frequent and severe transient fever and rigors, shortness of breath, and hypotension with rituximab. When these side effects are noted, the antibody infusion should be temporarily slowed or discontinued, the patient should be observed, and the severity of the side effects should be evaluated. The patient should be treated according to the best available local practices and procedures. Following observation, when the patient's symptoms improve, the infusion should be continued, initially at 1/2 the previous rate and gradually escalated to a maximum rate of 300 mg/hour (see table below). Subsequent infusions may be carried out at a gradually increased infusion rate of up to 400 mg/hr maximum. If the first dose of rituximab

is well tolerated, the starting flow rate for the administration of subsequent doses will be 100 mg/hr then increased gradually.

Following the antibody infusion, the IV line should be kept open for medications, as needed. If there are no complications, the IV line may be discontinued after one hour of observation. If complications occur during the rituximab infusion, the patient should be observed for two hours after the completion of the infusion.

| - | | | | | Mucosal | | |
|---|---|---|---|---|---|---|---|
| | | | | | congestion/ | | Drop in |
| Dose Rate | <u>Fever</u> | or | <u>Rigors</u> | or | <u>Edema</u> | or | <u>Systolic BP</u> |
| Decrease to 1/2 | > 38.5°C | | Mild | | Mild | | > 30 mm Hg |
| | | | Moderate | | Moderate | | 0 |

- 5.4.3 Adverse Clinical Events see Appendix E
- 5.5 Prophylaxis for Pneumocystis Carinii
  - 5.5.1 all patients will receive prophylaxis with trimethoprim-sulfa (TMP/SMX) as follows:

    Two DS tablets twice weekly on Saturday and Sunday.
  - 5.5.2 for TMP/SMX allergy, patients will receive pentamidine aerosol therapy: 300 mg q 4 weeks using a Respigard II neubulizer
  - 5.5.3 for any problems, please consult PI and/or ID
- 5.6 Dose Modification Guidelines
  - 5.6.1 Recommended Guidelines for Hematological Toxicity

| Lowest granulocyte | Lowest platelet | Modification |
|---|---|---|
| > 1000 and | >100,000 | Increase one level |
| >200 but <1000 or<br><200 for ≥ days | >20,000 but<br><100,000 | No change |
| <200 for > 5 days and/or | <20,000 | Decrease one level |
| Documented infection with neutropenia | Mucosal bleeding | Decrease one level |

5.6.2 For All Other Toxicities (see Appendix D)

Grade 0-2 No Change

- 3 Decrease one level
- 4 Stop Treatment

- 5.6.3 All courses will be held pending hematologic recovery to granulocytes >1,000 and platelets >100,000, and non-hematologic toxicities to grade <1.
- 5.6.4 Dose levels for FND

| <u>Level</u> | <u>-2</u> | <u>-1</u> | <u>0</u> | <u>+1</u> |
|------------------------|-----------|-----------|----------|-----------|
| Fludarabine (qd x 3) | $16/m^2$ | $20/m^2$ | $25/m^2$ | $30/m^2$ |
| Mitoxantrone (d.1) | $6.4/m^2$ | $8/m^2$ | $10/m^2$ | $12/m^2$ |
| Dexamethasone (qd x 5) | 20 mg | 20 mg | 20 mg | 20 mg |

- 5.7 Interferon alfa-2b (Intron A) Maintenance
  - 5.7.1 After completion of FND ± rituximab, patients will receive interferon alfa-2b (Intron A) maintenance.
  - 5.7.2 Maintenance (for CR, PR, and "CRu" patients)

| | day | 1 | 2 | 3 | 4-14 | |
|---|---|---|---|---|---|---|
| Dexamethasone (mg) | | 8 | 8 | 8 | - ) | Repeat q mo |
| Interferon (x $10^6$ u/m <sup>2</sup> ) | | 3 | 3 | 3 | 3 } | for 12 cycles |

5.7.3 IFN maintenance schedule for these receiving rituximab adjuvant therapy on delayed anti-CD20 arm:.

The IFN will start 1 month after the final FND course. Usually this will be before 12 months, i.e., <u>before</u> rituximab maintenance for patients on the delayed anti-CD20 arm.

When IFN and rituximab are given in the same month, the schedule will be as follows (see also 5.2.3):

| | day | 1 | 2+ | 3 | 4-15 |
|---|---|---|---|---|---|
| rituximab (mg/m²) | | 375 | - | - | - |
| dexamethasone (mg) | | 8* | 8 | 8 | - |
| Interferon alfa (x 10 <sup>6</sup> u/m <sup>2</sup> ) | | - | 3 | 3 | 3 |

<sup>\*</sup> decadron pre-med is optional but encouraged

#### 5.7.4 Dose Modification Guidelines for Interferon

| <u>Level</u> | <u>-2</u> | <u>-1</u> | <u>0</u> | <u>+1</u> |
|---|---|---|---|---|
| Interferon (x 10 <sup>6</sup> u/m <sup>2</sup> ) | 1 | 2 | 3 | 5 |

<sup>+</sup> day 2 if possible, but delay of 1-2 days permitted between rituximab and IFN

Interferon guidelines for hematologic toxicity same as for chemotherapy (see 5.6.1). For non hematologic toxicity:

#### Grade

- 0-1 Increase 1 level if appropriate (escalation anticipated to be done <u>infrequently</u>)
- 2 No change
- 3 Decrease 1 level
- 4 Hold treatment; discuss with study chairman

#### 6.0 PRETREATMENT EVALUATION (SEE APPENDIX A)

- 6.1 A complete history and physical to include performance status, recent weight loss, current weight and concurrent non-malignant disease and therapy. Detailed information on existing malignant lesions and sizes is required, within 2 weeks before starting therapy.
- 6.2 Laboratory studies shall include a CBC, platelet count, differential, urinalysis, chest x-ray, creatinine, electrolyte, bilirubin, SGOT, alkaline phosphate, and peripheral blood lymphocyte surface markers, LDH, assay for soluble CD20 if possible, and B2 microglobulin levels, to be done within 2 weeks before starting therapy.
- 6.3 Appropriate studies should be obtained to define fully the extent of disease. Bilateral bone marrow biopsy, chest x-ray and CAT scan of the area(s) of involvement should be performed within 2 months before therapy (within 1 month preferably, especially if there is any clinical evidence of rapidly changing adenopathy). Lymphangiogram is recommended but is optional. The measurements of masses detected by CT scan ideally should be recorded as the volume in cubic centimeters, or as the perpendicular diameters. All other masses should be recorded as the perpendicular diameter.
- 6.4 Baseline blood and bone marrow aspirates will be obtained for bcl-2 PCR. Contact our research nurse to make these arrangements, at the same time that eligibility screening is done. Please make these contacts early, so that candidate patients can have these studies done in a timely and efficient manner.
- 6.5 Immunophenotyping and gene rearrangement studies (PCR studies for bcl-2 mbr and mcr; and JH for bcl-2 negative patients) also should be performed on lymph node tissue, whenever possible. For fresh tissue obtained here, please arrange, through our research nurse, to have the sample triaged appropriately.

For biopsies done outside, prior to referral here, please arrange, through our research nurse, to have this archival tissue analyzed by Dr. Mederios.

For cases whose diagnosis is based on limited tissue sample (e.g., FNA), it is strongly encouraged to obtain more tissue. Please discuss such cases with the P.I., if it is felt that treatment plans need to proceed despite suboptimal diagnostic material.

- If fresh tissue is obtained, please also perform nucleic acid flow cytometry, if possible.
- 6.6 Required tests include ejection fraction by echocardiography or MUGA to be performed as baseline. Smokers as well as those with any significant history of pulmonary disease should also have pulmonary function testing. These should be done within 3 months before starting therapy.
- 6.7 Location, type and size of all measurable or evaluable lesions must be recorded prior to treatment.

#### 7.0 EVALUATION DURING STUDY (SEE APPENDIX A)

- 7.1. Patients shall be followed at least weekly with CBC, platelet count and differential and will be seen in our clinic after the second and fourth courses.
- 7.2 PCR in the peripheral blood will be followed every 6 months during the first 3 years, then every 12 months. PCR in the bone marrow will be followed every 6 months during the first 3 years, and every 12 months subsequently. For patients who are positive at the 6 month time point an additional PCR assay at 9 months is requested. For such patients who are still positive at 9 months, but who are subsequently negative at 12 months, yet another additional assay at 15 months is requested.
- 7.3 An SMA-12 shall be performed at least every other course or as frequently as needed to define drug toxicity.
- 7.4 Peripheral blood lymphocyte surface markers and Ig's every 3 months during therapy, and at least every 6-12 months off therapy until any abnormalities resolve.
- 7.5. Appropriate restaging every 3 courses, to include at least CXR, CT abdomen and pelvis, and BM Bx, and other tests to assess baseline measurable and assessable disease sites.
- 7.6 Cardiac re-evaluation as clinically indicated.
- 7.7 Off therapy monitoring should include restaging assessments (as outlined in section 7.5) at least every 6 months until relapse, or through year 5, and at least yearly thereafter.

#### 8.0 CRITERIA FOR RESPONSE AND TOXICITY

### 8.1 Tumor Measurements

a. Lesions will be measured bidimensionally in centimeters prior to each course of therapy. Masses detected by CT may be measured volumetrically in cubic centimeters.

- b. The longest diameter and its perpendicular will be measured on bidimensionally measured lesions. Size will be reported as the product of the diameters.
- c. Measurements should be made by the radiologist and/or clinician and recorded by the oncology research nurse under his/her supervision.
- d. An estimate of overall objective and subjective response will be made and recorded at each visit.

#### 8.2 Response Definitions:

- I. A molecular complete remission is defined as a patient with an initially positive peripheral blood PCR who converts to negative on at least 2 consecutive occasions no less than 2 months apart. If, during the interval when 2 consecutive blood PCR's are negative, a marrow PCR is positive, such patients would not be considered a molecular complete responder. (Such cases of discordance are infrequent but can occur).
- II. Clinical CR: defined as those who achieve a normal state which includes no detectable evidence of disease on x-rays.
- III. Clinical CRu: defined as "CR unconfirmed" on the basis of minimal residual abnormalities on x-ray such as a residual mass <25% of original measurement (either by volume calculation or by the product of 2 diameters -- See Sect. 8.1) with no palpable disease on physical examination.
- IV.Clinical PR: a) 50-75% reduction in the product of palpable tumor diameters of in the tumor volume measurements by radiologic criteria (See Sect. 8.1) or any palpable disease such as peripheral node(s) > 1 cm in diameter or palpable abdominal mass with histological evidence of lymphoma cells.
- V. Clinical minor response or failure includes, <50% tumor shrinkage or > 50%, but with tumor regrowth between courses.
- 8.3 All toxicities encountered during the study will be evaluated according to the grading system (0-4) in Appendix D and recorded prior to each course of therapy. Duration and treatment will be recorded. Life-threatening toxicities should be reported immediately to the Study Chairman.

#### 9.0 CRITERIA FOR REMOVAL FROM THE STUDY

- 9.1 Minor responses or failures to respond after delivering the first 4 courses of treatment in this protocol will be removed from the study.
- 9.2 Patients who relapse after achieving remission will be considered for ABMT or if not eligible will be treated with he salvage protocol of highest priority.

#### 10.0 STATISTICAL CONSIDERATIONS

10.1 Design:

The study will consist of a randomized controlled trial comparing two schedules of the anti-CD20 antibody rituximab, integrated with an established effective front-line chemotherapy program, FND. The primary endpoint will be the molecular complete response rate 12 months after the start of treatment. Since molecular response requires 2 consecutive negative PCR's (see 8.2, part I), a 12-month negative PCR will be considered truly negative only if a 9 or 15 month (or both) are also negative.

#### 10.2 Accrual Rate:

The average yearly accrual rate during the past 4 years on the current low grade lymphoma stage IV clinical trial has been 33 patients per year. Previous experience at M.D. Anderson Hospital has shown that the PCR positivity rate in these stages is in the neighborhood of 60% when tested with the mbr probe only. If the mcr probe is added, approximately 75% of patients can be expected to have a positive PCR at the time of diagnosis. Accrual of the target 128 evaluable patient (see 10.3 e) will therefore take just over 5 years (estimated 5 years, 2 months). Allowing for some inevaluable cases (9% on protocol 88-050), a total accrual of about 185 patients is planned. [Amendment May 2001: Planned accrual changed to 210 patients, with restriction of eligibility to follicular lymphoma only for the last 25-30 patients, so that adequate numbers are entered to fulfill the goal outlined in 10.3.a below. This amendment results from higher-than-expected numbers of patients with small lymphocytic (including MALT) lymphoma being entered.]

10.3 Adequacy of Sample Size:

Preliminary experience with the intensive regimen (CHOD-B/ESHAP/NOPP) has shown that a molecular CR rate in the neighborhood of 60-65% can be expected. Preliminary evidence indicates that a similar fraction of patients achieve molecular CR with FND.

An additional impact of rituximab is anticipated, since rituximab, when used singly, is capable of achieving blood and marrow molecular response, and rituximab has been integrated with CHOP chemotherapy with attainment of more molecular responses than would be expected with CHOP alone. Both the rapidity of attaining PCR-negative status, and the durability of the PCR-negative state, are additional molecular endpoints of interest. Thus, we intend to address if:

- a. the addition of biotherapy with chimeric anti-CD20 antibody to FND chemotherapy can induce a higher molecular response rate at 12 months than FND alone. This is the primary endpoint of this trial. The delayed administration of anti-CD20 given after 12 months, as in arm #1, will allow us to investigate this point. Sixty-four PCR-positive patients would be required in each arm to detect a difference of 25% in the 12-month molecular CR rates, assuming that the higher response rate was 85%. This assumes a two-sided  $\alpha$  level of 0.05 and a power of 0.90.
- b. the addition of biotherapy with anti-CD20 to FND chemotherapy (arm #2) is capable of inducing a higher molecular response rate at 6 months, as well as the 12 month primary endpoint, when compared with FND chemotherapy alone (arm #1).

- c. the addition of delayed anti-CD20 biotherapy after 12 months will then raise the molecular response rate at 18 months as compared with 12 months in the same patient. We will also compare the molecular response at 18 months with patients randomized to arm #2 (concurrent therapy) at the same timepoint.
- d. either of the two arms is associated with a more prolonged or sustained molecular response (as measured at 2 years from initiation of chemotherapy).
- e. the FFS of patients in the concurrent arm is different from the delayed arm. This is the secondary efficacy endpoint for which we can expect information on a reasonable time frame. (For survival, long-term follow-up is intended, but mature data requires 5-10 years follow-up -- which serves to emphasize the need to identify reliable surrogate endpoints). A 3-year FFS of 50% with standard therapy is typical. Assuming one FND plus rituximab scheme matches this standard expectation, and the other exceeds it by 20%, the trial will have power of 0.66 to detect a difference of this size at significance level of 0.05. This assumes that 128 patients will be entered at the rate of two patients per month, that FFS is distributed exponentially, and that all patients will be followed for a minimum of one year. Nonetheless, this data will: (a) be an important endpoint to correlate with the molecular remission data; and (b) hopefully provide hypothesis-generating information for future, larger-scale trials.

#### 10.4 Other Statistical Considerations

- a) Another secondary aim is to compare response rates, both CR (clinical CR plus CRu -- see Section 8.2) and CR + PR. It is anticipated to be high (approximately 80% CR and >90% CR + PR) in both arms; therefore it is unlikely that there will be significant differences between arms.
- b) Molecular response rates will be compared to CR and CR + PR rates.
- c) Other secondary aims, which are to compare the 5 year disease-free survival and overall survival for these 2 treatments, and to correlate the molecular complete remission rate with these endpoints, will require longer follow up. To attain these goals, we will follow the patients for at least 5 years to determine if a difference develops in disease-free survival. It might take 10 years or more of follow-up to establish statistically significant survival trends.
- d) Patients who are PCR negative will also be entered in this trial. These are of 2 categories: (a) "germline" follicular lymphoma; and (b) DSL (i.e., not follicular lymphoma).

Our preliminary data indicates that "germline" follicular patients have not done as well with FND as with ATT, so they will receive ATT, with rituximab. This will be a small number of patients (about 15% of follicular patients, i.e., about 16 patients on DM92-103), for whom analysis will be mainly descriptive. Likewise for DSL, which also will be a small subset of patients (24 in 4 1/2 years on DM92-103), traditional endpoints, including CR, PR, FFS, and survival will be used.

#### 11.0 DATA AND PROTOCOL MANAGEMENT

- 11.1 Protocol Compliance: The attending physician and oncology research nurse must see each patient at least every 2-3 cycles. All required interim and pretreatment data should be available and the physician must have made a designation as to tumor response and toxicity grade.
- 11.2 Data Entry: Data must be entered into the Clinical Data Management System. A brief explanation for required but missing data should be recorded as a comment.
- 11.3 Accuracy of Data Collection: The Study Chairman will be the final arbiter of response of toxicity should a difference of opinion exist.

### 12.0 REPORTING REQUIREMENTS

12.1 Any life-threatening and/or unexpected and serious (Grade 3 or 4) toxicity will be reported immediately to the Study Chairman who, in turn, must notify the Surveillance Committee and the sponsoring agency. Genentech Judith Canham 650-225-1000 x2330, Fax 650-225-4101.

#### 13.0 REFERENCES:

- 1. Rosenberg et al. Cancer 1982; 49:2112
- 2. Harris et al. Blood 1994; 84:1361
- 3. Fisher et al. Blood 1995; 85:1075
- 4. Martin et al. Blood 1995; 85:3671
- 5. WC Pugh personal communication
- 6. McLaughlin et al. In: Cabanillas & Rodriguez (eds) Advances in Lymphoma Research
- 7. Lopez-Guillermo et al. Blood 1996;88(Suppl 1): 34a
- 8. Horning. Semin Oncol 1993; 20:75
- 9. Jones et al. Cancer 1983; 51:1083
- 10. McLaughlin et al. In: Newland, Burnett, Keating, Armitage (eds) <u>Haematological</u> Oncology, Volume 1
- 11. McLaughlin. Biomed & Pharmacother 1996; 50:140
- 12. McLaughlin et al. Ann Oncol 1996; 7 (Suppl 3):34
- 13. McLaughlin et al. Ann Oncol 1994; 5 (Suppl 2):73
- 14. Lee, MŠ et al. Science 1987; 237:175
- 15. Gribben et al. NEJM 1991; 325:1525
- 16. Johnson et al. JCO 1994; 12:798
- 17. Lee MS. Semin Hematol 1993; 30:297
- 18. Lee MS et al. Blood 1988; 72(Suppl 1):247a
- 19. Gribben et al. Blood 1993; 81:3449
- 20. Cabanillas et al. Proc ASCO 1993; 12:365
- 21. Grossbard et al. Blood 1992; 80:863
- 22. Maloney et al. Blood 1994; 87:2457
- 23. McLaughlin et al. Blood 1996; 88 (Suppl 1):90a
- 24. Czuczman et al. Blood 1996; 88 (Suppl 1):453a
- 25. Demidem et al. Cancer Biother Radiopharm 1997; 12: 177
- 26. Cabanillas et al. Blood 1996; 88 (Suppl 1): 91a

#### APPENDIX A

#### **ACTIVITY FLOW CHART**

| | | | EVERY | EVERY | EVERY | |
|---|---|---|---|---|---|---|
| | PRE | | 2 | 3 | 6 | POST- |
| | STUDY | WEEKLY | COURSES | COURSES | MONTHS | THERAPY |
| H & P | X | | X | | | q 3-6 mo |
| PS | X | | | | | |
| CBC | X | X | | | | q 3-6 mo |
| U/A | X | | | | | |
| CXR | X | | | | | q 3-6 mo <sup>‡</sup> |
| SMA 12, K, MG* | X | | X | | | q 3-6 mo |
| B2M | X | | | X | | q 3-6 mo |
| BX/FNA* | X | | | | | |
| BM BX | X | | | X | | q 6 mo <sup>‡</sup> |
| LAG, CTs | X | | | X | | q 6 mo <sup>‡</sup> |
| PB markers, Ig's | X | | | X*** | | |
| PB PCR | X | | | | X** | |
| BM PCR | X | | | | X** | |
| ECHO or MUGA | X | | | | | |

- \* K, Mg, etc as indicated, mainly for pts on ATT (see App. B)
- \* when accessible; for phenotype, gene rearrangement
- \*\* PCR for bcl-2 q 6 mo yr 1-3, q 12 mo thereafter. Contingency for PCR monitoring at 9 and/or 15 months for selected patients (see 7.2)
- \*\*\* PB markers, Ig's: until recovery to normal
- ‡ Restaging off therapy (see section 7.7): at least q 6 mo until relapse or through year 5; then at least yearly.

#### APPENDIX B

MANAGEMENT STRATEGY FOR FOLLICULAR LYMPHOMA PATIENTS WHO DO NOT HAVE BCL-2 MBR OR MCR GENE REARRANGEMENT ("GERMLINE" PATIENTS).

I. Since these patients appear to have an inferior outcome with FND compared courses to ATT, these patients will receive ATT, 9 courses total, and all will also receive rituximab, 6 doses total. This will include d.1 and 8 doses of rituximab during the first cycles of CHOD-Bleo and NOPP (but not ESHAP) courses, and d.1 only during the second cycles of CHOD-Bleo and NOPP.

All "germline" patients will also receive interferon maintenance, as outlined for FND + rituximab patients (see 5.7).

Since the bcl-2 status may not be available prior to starting therapy, some will have received one (or rarely two) cycles of FND, with or without rituximab, prior to crossover to ATT. In such cases, the final chemotherapy cycle of the ATT sequence (NOPP) will be omitted, so that the total number of chemotherapy cycles is nine.

If the patient had been randomized to receive FND + rituximab and thus already received doses of rituximab, the subsequent courses of ATT, with d.1 and 8 IDEC during each CHOD-Bleo and NOPP course, should complete all 6 planned doses of rituximab (see scenario B below). For any patient who does <u>not</u> complete nine courses of chemotherapy, any missed doses of rituximab can be completed after the last chemotherapy cycle.

If the patient had been randomized to receive FND without rituximab, see scenario C.

#### Scenarios:

A. When the bcl-2 status is known before therapy (i.e., those patients who are not randomized -- see section 5.1.1):

course 1: CHOD-Bleo, plus rituximab d. 1 & 8

course 2: ESHAP

course 3: NOPP, plus rituximab d.1 & 8

course 4: CHOD-Bleo, plus rituximab d.1 only

course 5: ESHAP

course 6: NOPP, plus rituximab d.1 <u>only</u>

courses 7-9: CHOD-Bleo; ESHAP; NOPP (No more rituximab)

B. If patient had been randomized, and got FND with rituximab:

course 1: FND + rituximab d. 1 & 8

course 2: CHOD-Bleo, plus rituximab d.1 & 8

course 3: ESHAP

course 4: NOPP, plus rituximab d.1 & 8

course 5: CHOD-Bleo without rituximab

course 6: ESHAP

courses 7-9: NOPP; CHOD-Bleo; ESHAP (No more rituximab)

# C. If patient had been randomized, and got FND without rituximab:

course 1: FND

course 2: CHOD-Bleo, plus rituximab d. 1 & 8

course 3: ESHAP

course 4: NOPP, plus rituximab d. 1 & 8

course 5: CHOD-Bleo, plus rituximab d. 1 & 8

course 6: ESHAP

courses 7-9: NOPP; CHOD-Bleo; ESHAP (no more rituximab)

For any questions about this sequence, consult P.I.

For all cycles given in conjunction with rituximab, the steroid will start on d. 1 along with the rituximab, and the remainder of the chemotherapy will start one day later than standard, analogous to the modified schedule of FND as outlined in Section 5.

## II. ATT doses and schedule (with rituximab in CHOD-Bleo and NOPP courses):

## 1. Initial Dosing Regimen for CHOD-Bleo:

| Agent | <u>Dose</u> | <u>Days</u> | Route | <u>Time</u> | Total Dose |
|---|---|---|---|---|---|
| Rituximab | $375 \mathrm{mg/m^2}$ | 1 & 8 | IV | approx 4 hr | 750 mg/m <sup>2</sup> |
| | | | | (Sec 5. 4) | |
| Adriamycin | 25 mg/m²/day | 2-3 | IV-CI | 48 hrs | $50 \text{mg/m}^2$ |
| Oncovin | $0.7 \mathrm{mg/m^2/day}$ | 2-3 | IV-CI | 48 hrs | $1.4 \mathrm{mg/m^2}$ |
| Bleomycin | 5 u/m²/day | 2-3 | IV-CI | 48 hrs | $10 \text{ u/m}^2$ |
| Cytoxán | 750 mg/m <sup>2</sup> | 2 | IVPB | 15 min | 750 mg/m² |
| Dexamethasone | 40 mg/day | 1-4 | p.o. | | 160 mg |

## 2. Initial Dosing Regimen for ESHAP:

| Agent<br>Etoposide | $\frac{\text{Dose}}{40 \text{ mg/m}^2}$ | <u>Days</u><br>1-4 | Route<br>IV | <u>Time</u><br>30 min | Total Dose<br>160 mg/m <sup>2</sup> |
|---|---|---|---|---|---|
| • | (daily)<br>25 mg/m <sup>2</sup> | 1-4 | IV-CI | 96 hrs | $100 \mathrm{mg/m^2}$ |
| Cisplatin | (daily) | | | | <u>.</u> |
| Ara-C | 1.5 gm/m <sup>2</sup> (single dose) | 5 | IV | 2 hrs | $1.5 \mathrm{gm/m^2}$ |
| Solu Medrol | 500 mg<br>(daily) | 1-5 | IV | 15 min | 2500 mg |

## 3. Initial Dosing Regimen for NOPP:

| _ | - | | | | |
|---|---|---|---|---|---|
| Agent | Dose | Days | Route | Time approx 4 hr | Total Dose |
| Rituximab | 375 mg/m² | 1 & 8 | IV | | 750 mg/m² |
| Novantrone | 10 mg/m²<br>(single dose) | 2 | IV | (Sec 5.4)<br>15 min | $10\mathrm{mg/m^2}$ |
| Oncovin | 1.4 mg/m <sup>2</sup> | 2 | IVPB | 15 min | 1.4 mg/m <sup>2</sup> |
| Procarbazine | 100 mg/m <sup>2</sup> | 2-11 | p.o. | | 1000 mg/m <sup>2</sup> |
| Prednisone | 100 mg | 1-5 | p.o | | 500 mg |

# III. Dose modifications related to myelotoxicity.

# 1. For CHOD-Bleo

| Dose Level: | -2 | -1 | 0 | 1 |
|---|---|---|---|---|
| Adriamycin<br>( <u>total</u> dose) | $35 \mathrm{mg/m^2}$ | 40 mg/m <sup>2</sup> | $50 \mathrm{mg/m^2}$ | $60 \text{ mg/m}^2$ |
| Cytoxan | $500 \text{ mg/m}^2$ | $600 \text{mg/m}^2$ | $750 \text{ mg/m}^2$ | $1000 \text{ mg/m}^2$ |
| Oncovin<br>( <u>total</u> dose) | $1.4 \text{ mg/m}^2$ | $1.4 \text{ mg/m}^2$ | $1.4 \mathrm{mg/m^2}$ | $1.4 \text{ mg/m}^2$ |
| Bleomycin<br>( <u>total</u> dose) | 10 u/m² | 10 u/m <sup>2</sup> | $10 \text{ u/m}^2$ | 10 u/m <sup>2</sup> |
| Dexamethasone (daily dose) | 40 mg | 40 mg | 40 mg | 40 mg |
| 2. For ESHAP | | | | |
| Dose Level: | <u>-2</u> | -1 | 0 | 1 |
| Etoposide<br>(daily dose) | 25 mg/m <sup>2</sup> | $30 \text{ mg/m}^2$ | $40 \text{ mg/m}^2$ | $50 \text{ mg/m}^2$ |
| Cisplatin<br>(daily dose) | 16 mg/m <sup>2</sup> | $20 \text{ mg/m}^2$ | $25 \text{ mg/m}^2$ | 25 mg/m <sup>2</sup> |
| Ara-C x1 | $0.5 \mathrm{mg/m^2}$ | $1 \text{ g/m}^2$ | $1.5 \mathrm{mg/m^2}$ | $2 g/m^2$ |
| Solu Medrol<br>(daily dose) | 500 mg | 500 mg | 500 mg | 500 mg |
| 3. For NOPP<br>Dose Level: | -2 | -1 | 0 | 1 |
| Novantrone | 6 mg/m <sup>2</sup> | 8 mg/m <sup>2</sup> | $10 \text{mg/m}^2$ | $12 \text{mg/m}^2$ |
| Oncovin | $1.4 \text{ mg/m}^2$ | $1.4 \mathrm{mg/m^2}$ | $1.4\mathrm{mg/m^2}$ | $1.4 \text{ mg/m}^2$ |
| Procarbazine<br>(daily dose) | 60 mg/m <sup>2</sup> | 80 mg/m <sup>2</sup> | $100 \text{ mg/m}^2$ | 120 mg/m <sup>2</sup> |
| Prednisone<br>(daily dose) | 100 mg | 100 mg | 100 mg | 100 mg |

# IV. Recommended Dose Modification Guidelines

For Hematologic Toxicity -- see Section 5.6
 For Renal Toxicity

| Serum Creat<br>(mg%) | inine | Creatinine Clearance<br>(cc/min) | Modification of Cisplatin |
|---|---|---|---|
| 0.6 - 1.4 | or | > 75 | None |
| 1.5 - 2.0 | or | 60 - 74 | 33% reduction |
| 2.1 - 2.5 | or | 40 - 59 | 50% reduction |
| >2.5 - 4.0 | or | <39 | Delete* |

<sup>\*</sup> Cisplatin could be given at 25% dose, after consultation with Study Chairman, if renal failure is secondary to lymphoma.

#### APPENDIX C

#### PERFORMANCE STATUS SCALES

## Karnofsky Performance Scale (1)

### Zubrod Performance Scale (2)

| Point | Description | Point | Description |
|---|---|---|---|
| 100 | Normal, no complaints, no evidence of disease | 0 | Normal activity; asymptomatic |
| 90 | Able to carry on normal activity; minor signs or symptoms of disease | 1 | Symptomatic; but ambulatory |
| 80 | Normal activity with effort; some signs or symptoms of disease | | · |
| 70 | Cares for self, unable to carry on normal activity or to do active work | 2 | Symptomatic; in bed 50% of time |
| 60 | Requires occasional assistance, but able to care for most of own needs | | |
| 50 | Requires considerable assistance and frequent medical care | 3 | Symptomatic; in bed<br>50% of time; not<br>bedridden |
| 40 | Disabled, requires special care and assistance | | |
| 30 | Severely disabled, hospitalization indicated. Death not imminent | 4 | 100% bedridden |
| 20 | Very sick, hospitalization indicated. Death not imminent | | |
| 10 | Moribund, fatal processes, progressing rapidly | | |
| 0 | Dead | 5 | Dead |

#### **REFERENCES**

- 1. Karnofsky, D.A: Meaningful Clinical Classification of Therapeutic Responses to Anti-Cancer Drugs. Editorial. <u>Clin. Pharmacol and Therapeutics</u> 2:709-712, 1961.
- 2. Stanley, K.E.: Prognostic Factors for Survival in Patients with Inoperable Lung Cancer. <u>J. Natl. Can. Inst.</u> 65:25-32, 1980.

# APPENDIX D

# NCI COMMON TOXICITY CRITERIA

| | | Grade | C | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | ALLERGY/IMM | UNOLOGY | | |
| Allergic reaction/<br>hypersensitivity<br>(including drug<br>fever)<br>Note: Isolated urticaria | none<br>n, in the absence | transient rash,<br>drug fever <<br>38°C (<100.4°F)<br>e of other manifestation | urticaria, drug fever ≥ 38°C (≥100.4°F), and/or asymptomatic bronchospasm | symptomatic<br>bronchospasm,<br>requiring<br>parenteral<br>medication(s),<br>with or without<br>urticaria; allergy-<br>related<br>edema/angioede<br>ma<br>persensitivity reaction | anaphylaxi |
| graded in the DERMA | | | moderate, | - | - |
| Allergic rhinitis<br>(including sneezing,<br>nasal stuffiness,<br>postnasal drip) | none | mild, not<br>requiring<br>treatment | requiring<br>treatment | | |
| Autoimmune | none<br>yroidism, Colit | serologic or other evidence of autoimmune reaction but patient is asymptomatic (e.g., vitiligo), all organ function is normal and no treatment is required | evidence of autoimmune reaction involving a non- essential organ or function (e.g., hypothyroidism), requiring treatment other than immunosuppress ive drugs | reversible autoimmune reaction involving function of a major organ or other toxicity (e.g., transient colitis or anemia), requiring short- term immunosuppress ive treatment | autoimmure reaction causing major grad 4 organ dysfunction progressive and irreversible reaction; long-term administra on of high-dose immunosuppressive therapy required |
| Serum sickness | none | _ | - | present | - |
| Urticaria is graded in to other manifestations of | the DERMATO<br>f allergic or hy | DLOGY/SKIN category<br>persensitivity reaction, | rit it occurs as an isol<br>, grade as Allergic rea | ated symptom. If it o<br>action/hypersensitiv | occurs with<br>ity above. |
| Vasculitis | none | mild, not<br>requiring<br>treatment | symptomatic,<br>requiring<br>medication | requiring<br>steroids | ischemic<br>changes or<br>requiring<br>amputation |
| Allergy/Immunolog<br>y-Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disablin |
| / | | AUDITORY/I | HEARING | | |
| | | Middle ear/hearing ir | | | |

| | | Grade | | | _ |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Earache is graded in the External auditory canal Note: Changes associat | normal ed with radiation | external otitis with erythema or dry desquamation | external otitis<br>with moist<br>desquamation<br>nae) are graded unde | external otitis<br>with discharge,<br>mastoiditis<br>er Radiation dermatit | necrosis of<br>the canal<br>soft tissue<br>or bone<br>is in the |
| DERMATOLOGY/SKI | | hearing loss on | tinnitus or | tinnitus or | severe |
| Inner ear/hearing | normal | audiometry only | hearing loss, not<br>requiring hearing<br>aid or treatment | hearing loss,<br>correctable with<br>hearing aid or<br>treatment | unilateral or<br>bilateral<br>hearing loss<br>(deafness),<br>not<br>correctable |
| Middle ear/hearing | normal | serous otitis<br>without<br>subjective<br>decrease in<br>hearing | serous otitis or infection requiring medical intervention; subjective decrease in hearing; rupture of tympanic membrane with discharge | otitis with<br>discharge,<br>mastoiditis or<br>conductive<br>hearing loss | necrosis of<br>the canal<br>soft tissue<br>or bone |
| Auditory/Hearing-<br>Other<br>(Specify, | normal | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | BLOOD/BONE | MARROW | | |
| Bone marrow cellularity | normal for<br>age | mildly<br>hypocellular or<br>25% reduction<br>from normal<br>cellularity for age | moderately hypocellular or >25 - ≤ 50% reduction from normal cellularity for age or >2 but <4 weeks to recovery of normal bone marrow cellularity | severely hypocellular or >50 - ≤ 75% reduction in cellularity for age or 4 - 6 weeks to recovery of normal bone marrow cellularity | aplasia or >6 weeks to recovery of normal bone marrow cellularity |
| Normal ranges:<br>children (≤ 18 years)<br>younger adults (19-<br>59) | 90% cellularity average 60-70% cellularity average | | , | | |
| older adults (≥ 60 years) | 50%<br>cellularity<br>average | | | | |
| Note: Grade Bone mar | row cellularity or<br>WNL | nly for changes relate<br>< LLN - | ed to treatment not d<br>200 - < 500/mm <sup>3</sup> | isease.<br>50 - < 200/mm <sup>3</sup> | < 50/mm <sup>3</sup> |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| <b>Foxicity</b> | 0 | 1 | 2 | 3 | 4 |
| Haptoglobin | normal | decreased | - | absent | - (1) |
| Hemoglobin (Hgb) | WNL | < LLN - 10.0 g/dl<br>< LLN - 100 g/L<br>< LLN - 6.2 | 8.0 - < 10.0 g/dl<br>80 - < 100 g/L<br>4.9 - < 6.2 | 6.5 - < 8.0 g/dl<br>65 - 80 g/L<br>4.0 - < 4.9 | < 6.5 g/dl<br>< 65 g/L<br>< 4.0 |
| | | mmol/L | mmol/L | mmol/L | mmol/L |
| Note: The following cr<br>If the protocol so speci | iteria may be use | d for leukemia studio | es or bone marrow i | nfiltrative/myelophth | usic process |
| If the protocol so speci<br>For leukemia studies<br>or bone marrow<br>infiltrative/<br>myelophthisic<br>processes | wnL | 10 - <25%<br>decrease from<br>pretreatment | 25 - <50%<br>decrease from<br>pretreatment | 50 - <75%<br>decrease from<br>pretreatment | ≥75%<br>decrease<br>from<br>pretreatmer<br>t |
| Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis, other) | none | only laboratory<br>evidence of<br>hemolysis [e.g.,<br>direct<br>antiglobulin test<br>(DAT, Coombs')<br>schistocytes] | evidence of red cell destruction and ≥ 2gm decrease in hemoglobin, no transfusion | requiring<br>transfusion<br>and/or medical<br>intervention (e.g.,<br>steroids) | catastrophic<br>consequenc<br>es of<br>hemolysis<br>(e.g., renal<br>failure,<br>hypotension |
| ., ., ., ., | Jahin II-la | | | | bronchospa<br>m,<br>emergency<br>splenectom<br>y) |
| Also consider Haptog | | < LLN - 3.0 x 10 <sup>9</sup> | $\geq 2.0 - < 3.0 \times 10^9$ | $\geq 1.0 - < 2.0 \times 10^9$ | < 1.0 x 10 <sup>9</sup> |
| Leukocytes (total<br>WBC) | WNL | /L<br>< LLN -<br>3000/mm <sup>3</sup> | /L<br>≥2000 - <<br>3000/mm³ | /L<br>≥1000 - <<br>2000/mm³ | /L<br>< 1000/mm |
| For BMT studies: | WNL | ≥2.0 - <3.0 X<br>10 <sup>9</sup> /L<br>≥2000 -<br><3000/mm <sup>3</sup> | ≥1.0 - <2.0 x 10°<br>/L ≥1000 -<br><2000/mm³ | ≥0.5 - <1.0 x 10°<br>/L ≥500 -<br><1000/mm³ | <0.5 x 10°<br>/L<br><500/mm³ |
| Note: The following crit | eria using age, rac | e and sex normal value | s may be used for pedi | atric studies if the proto | col so |
| specifies. | | ≥75 - <100% LLN | ≥50 - <75% LLN | ≥25 - 50% LLN | <25% LLN |
| Lymphopenia | WNL | <lln -="" 1.0="" 10<sup="" x="">9 /L <lln -="" 1000="" mm<sup="">3</lln></lln> | ≥0.5 - <1.0 x 10 <sup>9</sup> /L ≥500 - <1000/mm <sup>3</sup> | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> | - |
| Note: The following crit | teria using age, rac | e, and sex normal valu | es may be used for ped | iatric studies if the prot | ocol so |
| specifies. | | ≥75-<100%LLN | ≥50-<75%LLN | ≥25-<50%LLN | <25%LLN |
| Neutrophils/granul | WNL | ≥1.5 - <2.0 x 10 <sup>9</sup> | ≥1.0 - <1.5 x 10 <sup>9</sup> | ≥0.5 - <1.0 x 10 <sup>9</sup> | < 0.5 x 10 <sup>9</sup><br>/L |
| ocytes<br>(ANC/AGC) | | /L<br>≥1500 -<br><2000/mm³ | /L<br>≥1000 -<br><1500/mm³ | /L<br>≥500 -<br><1000/mm³ | < 500/mm |
| For BMT: | WNL | ≥1.0 - <1.5 x 10 <sup>9</sup> /L ≥1000 - <1500/mm <sup>3</sup> | ≥0.5 - <1.0 x 10 <sup>9</sup> /L ≥500 - <1000/mm <sup>3</sup> | ≥0.1 - <0.5 x 10 <sup>9</sup><br>/L<br>≥100 - <500/mm <sup>3</sup> | <0.1 x 10 <sup>9</sup><br>/L<br><100/mm <sup>3</sup> |
| 4 ≥75% decrease from baseline 0 x < 10.0 x 10 /L < 10000/mm 1 x 109 < 10.0 x 109 |
|---|
| decrease from baseline 0 x < 10.0 x 10 /L < 10000/mm 0 x 109 < 10.0 x 109 |
| from baseline 0 x < 10.0 x 10 /L < 10000/mm 0 x 109 < 10.0 x 109 |
| baseline 0 x < 10.0 x 10 /L < 10000/mm 0 x 109 < 10.0 x 109 |
| 0 x < 10.0 x 100 /L < 100000/mm |
| /L<br><<br>10000/mm<br>× 10° <10.0 x 10° |
| /L<br><<br>10000/mm<br>× 10° <10.0 x 10° |
| <pre></pre> |
| 10000/mm<br>x 10 <sup>9</sup> <10.0 x 10 <sup>9</sup> |
| $\times 10^9 < 10.0 \times 10^9$ |
| /L |
| <10000/m |
| 3 3 |
| elophthisic process |
| stophulasic process |
| ≥75% |
| m decrease |
| from |
| baseline |
| baseine |
| .1.(.1.) |
| platelet<br>transfusion |
| and other |
| measures |
| required to |
| improve |
| platelet |
| increment |
| platelet |
| transfusio |
| refractorin |
| s associate |
| with life- |
| threatenin |
| bleeding. |
| (e.g., HĽA |
| or cross |
| matched |
| platelet |
| transfusion |
| ) |
| , |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| For BMT: | none | 1 platelet<br>transfusion in 24<br>hours | 2 platelet<br>transfusions in 24<br>hours | ≥3 platelet<br>transfusions in 24<br>hours | platelet<br>transfusions<br>and other<br>measures<br>required to<br>improve<br>platelet<br>increment;<br>platelet<br>transfusion<br>refractorines<br>s associated<br>with life-<br>threatening |
| | | | | | bleeding. |
| | | | | | (e.g., HLA |
| | | | | | or cross<br>matched<br>platelet<br>transfusions<br>) |
| Also consider Plate | | | | Yes | |
| Transfusion: pRBCs For BMT: Also consider Hem | none | ≤2 u pRBC<br>(≤15cc/kg) in 24<br>hours elective or<br>planned | 3 u pRBC (>15<br>≤30cc/kg) in 24<br>hours elective or<br>planned | Yes<br>≥4 u pRBC<br>(>30cc/kg) in 24<br>hours | hemorrhage<br>or<br>hemolysis<br>associated<br>with life-<br>threatening<br>anemia;<br>medical<br>intervention<br>required to<br>improve<br>hemoglobin |
| Blood/Bone | none | mild | moderate | severe | life- |
| Marrow-Other<br>(Specify, | 110110 | | | | threatening<br>or disabling |
| | | CARDIOVASCULAR | (ARRHYTHMIA) | | |
| Conduction<br>abnormality/<br>Atrioventricular<br>heart block | none | asymptomatic,<br>not requiring<br>treatment (e.g.,<br>Mobitz type I<br>second-degree<br>AV block,<br>Wenckebach) | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment (e.g.,<br>Mobitz type II<br>second-degree<br>AV block, third-<br>degree AV block) | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Nodal/junctional<br>arrhythmia/dysrhyt<br>hmia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| Palpitations<br>Note: Grade palpitation | none | present | -<br>d arrhythmia | - | - |
| Prolonged QTc interval (QTc > 0.48 seconds) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| Sinus bradycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| Sinus tachycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment of<br>underlying cause | - |
| Supraventricular arrhythmias (SVT/atrial fibrillation/ flutter) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| Syncope (fainting) is | | UROLOGY category. | 1 | | |
| Vasovagal episode | none | - | present without<br>loss of<br>consciousness | present with loss<br>of consciousness | - |

| | | Grade | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Ventricular<br>arrhythmia<br>(PVCs/bigeminy/tri<br>geminy/<br>ventricular<br>tachycardia) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| Cardiovascular/<br>Arrhythmia-Other<br>(Specify,<br>) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic,<br>and requiring<br>treatment of<br>underlying cause | life-<br>threatening<br>(e.g.,<br>arrhythmia<br>associated<br>with CHF,<br>hypotension<br>, syncope,<br>shock) |
| | | CARDIOVASCULA | R (GENERAL) | | |
| Acute vascular leak<br>syndrome | absent | - | symptomatic, but<br>not requiring<br>fluid support | respiratory<br>compromise or<br>requiring fluids | life-<br>threatening;<br>requiring<br>pressor<br>support<br>and/or<br>ventilatory<br>support |
| Cardiac-<br>ischemia/infarction | none | non-specific T-<br>wave flattening<br>or changes | asymptomatic,<br>ST- and T- wave<br>changes<br>suggesting<br>ischemia | angina without<br>evidence of<br>infarction | acute<br>myocardial<br>infarction |
| Cardiac left<br>ventricular function | normal | asymptomatic decline of resting ejection fraction of ≥ 10% but < 20% of baseline value; shortening fraction ≥ 24% but < 30% | asymptomatic but resting ejection fraction below LLN for laboratory or decline of resting ejection fraction ≥ 20% of baseline value; < 24% shortening fraction | CHF responsive<br>to treatment | severe or<br>refractory<br>CHF or<br>requiring<br>intubation |
| CNS cerebrovascular | ischemia is grad | ded in the NEUROLOG | GY category. | 1 | larvala |
| Cardiac troponin I<br>(cTnI) | normal | - | - | levels consistent<br>with unstable<br>angina as defined<br>by the<br>manufacturer | levels consistent with myocardial infarction as defined by the manufactur er |
| Cardiac troponin T (cTnT) | normal | ≥ 0.03 - < 0.05<br>ng/ml | $\geq 0.05 - < 0.1$ ng/ml | $\geq 0.1 - < 0.2$ ng/ml | ≥ 0.2 ng/ml |

| | | Grad | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Edema | none | asymptomatic,<br>not requiring<br>therapy | symptomatic,<br>requiring therapy | symptomatic edema limiting function and unresponsive to therapy or requiring drug discontinuation | anasarca<br>(severe<br>generalized<br>edema) |
| Hypertension | none | asymptomatic,<br>transient increase<br>by >20 mmHg<br>(diastolic) or to ><br>150/100* if<br>previously WNL;<br>not requiring<br>treatment | recurrent or<br>persistent or<br>symptomatic<br>increase by > 20<br>mmHg (diastolic)<br>or to > 150/100*<br>if previously<br>WNL; not<br>requiring<br>treatment | requiring therapy<br>or more intensive<br>therapy than<br>previously | hypertensiv<br>e crisis |
| | | sex appropriate normal changes, but not | values > 95th percentu<br>requiring brief | e ULN.<br>requiring therapy | shock |
| Hypotension | none | requiring therapy<br>(including<br>transient<br>orthostatic<br>hypotension) | fluid replacement<br>or other therapy<br>but not<br>hospitalization;<br>no physiologic<br>consequences | and sustained medical attention, but resolves without persisting physiologic consequences | (associated with acidemia and impairing vital organ function due to tissue hypoperfusion) |
| category. For pediatric paties | is graded as Ca<br>nts, systolic BP 6 | rdiac- ischemia/infarc<br>5 mmHg or less in infan<br>ve or three measurements | ts up to 1 year old and | | |
| Myocarditis | none | - | - | CHF responsive to treatment | severe or<br>refractory<br>CHF |
| Operative injury of<br>vein/artery | none | primary suture<br>repair for injury,<br>but not requiring<br>transfusion | primary suture<br>repair for injury,<br>requiring<br>transfusion | vascular<br>occlusion<br>requiring surgery<br>or bypass for<br>injury | myocardial<br>infarction;<br>resection of<br>organ (e.g.,<br>bowel, limb |
| Pericardial effusion/<br>pericarditis | none | asymptomatic<br>effusion, not<br>requiring<br>treatment | pericarditis (rub,<br>ECG changes,<br>and/or chest<br>pain) | physiologic<br>consequences<br>resulting from<br>symptoms | tamponade<br>(drainage of<br>pericardial<br>window<br>required) |
| Peripheral arterial<br>ischemia | none | - | brief episode of ischemia managed non-surgically and without permanent deficit | requiring<br>surgical<br>intervention | life-<br>threatening<br>or with<br>permanent<br>functional<br>deficit (e.g.,<br>amputation |

| | | Grad | le | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Phlebitis | none | - | present | • | - |
| (superficial) | | | 1 | | |
| Note: Injection site r | eaction is graded | d in the DERMATOL | OGY/SKIN category | • | |
| Thrombosis/emb | polism is graded | in the CARDIOVASO | CULAR (GENERAL) | category. | |
| Syncope (fainting) is g | raded in the NE | IROLOGY category. | / | | |
| Thrombosis/embolis | | - | deep vein | deep vein | embolic |
| · | Horie | | thrombosis, not | thrombosis, | event |
| m | | | requiring | requiring | including |
| | | | anticoagulant | anticoagulant | pulmonary |
| | | | artificoaguiarte | therapy | embolism |
| Vein/artery operative | iminum, in anadod | as Operative injury | of wain /artary in that | | |
| | | as Operative figury ( | or veni/artery ni nie v | CANDIOVASCOLAI | • |
| (GENERAL) category. | | | herial amissada of | un acciding | life- |
| Visceral arterial | none | - | brief episode of | requiring | |
| ischemia (non- | | | ischemia | surgical | threatening |
| myocardial) | | | managed non- | intervention | or with |
| | | | surgically and | | permanent |
| | | | without | | functional |
| | | • | permanent deficit | | deficit (e.g., |
| | | | | | resection of |
| | | | | | ileum) |
| Cardiovascular/ | none | mild | moderate | severe | life- |
| General-Other | | | | | threatening |
| (Specify, | | | | | or disabling |
| ) | | | | | |
| | | COAGUL | ATION | | |
| Note: See the HEMOR | RHAGE categor | y for grading the sev | erity of bleeding ever | nts. | |
| DIC | absent | - | • | laboratory | laboratory |
| (disseminated | | | | findings present | findings |
| intravascular | | | | with <u>no</u> bleeding | and |
| coagulation) | | | | | bleeding |
| Also grade Platelets. | | | | | Ü |
| Note: Must have incre | ased fibrin split | products or D-dimer | in order to grade as l | DIC. | |
| Fibrinogen | WNL | ≥0.75 - <1.0 x | ≥0.5 - <0.75 x | ≥0.25 - <0.5 x | <0.25 x LLN |
| | | LLN | LLN | LLN | |
| Note: The following c | riteria may be us | | | | hisic process |
| if the protocol so spec | | | | | 1 |
| For leukemia | WNL | <20% decrease | ≥20 - <40% | ≥40 - <70% | <50 mg% |
| studies: | MILL | from | decrease from | decrease from | . 100 22.670 |
| bradies. | | pretreatment | pretreatment | pretreatment | |
| | | value or LLN | value or LLN | value or LLN | |
| Partial | WNL | > ULN - ≤ 1.5 x | > 1.5 - ≤ 2 x ULN | >2 x ULN | |
| | AATAD | ULN | > 1.0 - 3 Z X OLIN | /Z A ULIN | • |
| thromboplastin time | | OFIA | | | |
| (PTT) | th a CADDIOVA | CCIII AD (CENTED AT | \ antogowy | | |
| Phelbitis is graded in | | | | . O TII NY | |
| Prothrombin time | WNL | > ULN - ≤ 1.5 x | $> 1.5 - \le 2 \times ULN$ | >2 x ULN | - |
| (PT) | , | ULN | ID (CITATED AT) | Market Commencer | |
| Thrombosis/embolism | n is graded in th | e CARDIOVASCULA | AK (GENEKAL) categ | ory. | |

| 0 | 4 | | | |
|---|---|---|---|---|
| | 1 | 2 | 3 | 4 |
| absent | | - | laboratory findings present without clinical consequences | laboratory findings and clinical consequenc es, (e.g., CNS hemorrhage / bleeding or thrombosis/ embolism or renal failure) requiring therapeutic intervention |
| | evidence of RBC<br>destruction<br>(schistocytosis)<br>without clinical<br>consequences | evidence of RBC destruction with elevated creatinine (≤3 x ULN) | evidence of RBC<br>destruction with<br>creatinine (>3 x<br>ULN) not<br>requiring dialysis | evidence of RBC destruction with renal failure requiring dialysis and/or encephalopa thy |
| lobin (Hgb), Plate | elets, Creatinine. | (e.g. schistocytes, he | elmet cells, red cell fr | agments). |
| none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| none | increased fatigue<br>over baseline, but<br>not altering<br>normal activities | moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or Lansky) or causing difficulty performing some activities | severe (e.g., decrease in performance status by ≥2 ECOG levels or 40% Karnofsky or Lansky) or loss of ability to perform some activities | bedridden<br>or disabling |
| | none none | destruction (schistocytosis) without clinical consequences lobin (Hgb), Platelets, Creatinine. oangiopathic changes on blood smear none mild CONSTITUTIONA none increased fatigue over baseline, but not altering | destruction (schistocytosis) elevated creatinine (≤3 x consequences ULN) lobin (Hgb), Platelets, Creatinine. coangiopathic changes on blood smear (e.g., schistocytes, he none mild moderate CONSTITUTIONAL SYMPTOMS none increased fatigue over baseline, but not altering normal activities moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or Lansky) or causing difficulty performing some activities | evidence of RBC destruction (schistocytosis) without clinical consequences Consequences Co |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Γoxicity | 0 | 1 | 2 | 3 | 4 |
| Pever (in the absence | none | 38.0 - 39.0°C | 39.1 - 40.0°C | > 40.0°C | > 40.0°C |
| of neutropenia, | 110110 | (100.4 - 102.2°F) | (102.3 - 104.0°F) | (>104.0°F) for < | (>104.0°F) |
| where neutropenia | | | | 24hrs | for > 24hrs |
| s defined as AGC < | | | | | |
| 1.0 x 10 <sup>9</sup> /L) | | | | | |
| Also consider Allergic | reaction / hyperse | nsitivity. | | | |
| Note: The temperature | measurements li | sted above are oral | or tympanic. | | |
| Hot flashes/flushes are | e graded in the El | NDOCRINE categor | v. | | |
| Rigors, chills | none | mild, requiring | severe and/or | not responsive to | - |
| rugors, crims | 110110 | symptomatic | prolonged, | narcotic | |
| | | treatment (e.g., | requiring | medication | |
| | | blanket) or non- | narcotic | | |
| | | narcotic | medication | | |
| | | medication | 11100120111011 | | |
| | | mild and | frequent or | - | - |
| Sweating | normal | occasional | drenching | | |
| (diaphoresis) | <b>PO</b> / | | 10 - <20% | ≥ 20% | - |
| Weight gain | < 5% | 5 <b>-</b> <10% | 10 - <20 /0 | ≥ 20 /0 | |
| Also consider Ascites, | Edema, Pleural e | frusion. | | | |
| (VOD)<br>Note: The following c | <2% | ≥2 - <5% | 25 - <10% | ascities | ≥10% or<br>fluid<br>retention<br>resulting in<br>pulmonary<br>failure |
| Weight loss | < 5% | 5 - <10% | 10 - <20% | ≥20% | |
| Also consider Vomitin | ng, Dehydration, | Diarrhea. | | | - |
| | | | | | - |
| Constitutional | none | mild | moderate | severe | life- |
| | none | | moderate | severe | threatening |
| Symptoms-Other | none | | moderate | severe | threatening |
| | none | | moderate | severe | life-<br>threatening<br>or disabling |
| Symptoms-Other | none | mild | ,, | severe | threatening |
| Symptoms-Other (Specify, | | mild DERMATOL | OGY/SKIN | severe | threatening |
| Symptoms-Other | none | mild | OGY/SKIN pronounced hair loss | | threatening |
| Symptoms-Other (Specify, Alopecia Bruising | | DERMATOL mild hair loss localized or in | OGY/SKIN pronounced hair | | threatening |
| Symptoms-Other (Specify, Alopecia Bruising (in absence of grade 3 or 4 | normal | mild DERMATOL mild hair loss | OGY/SKIN pronounced hair loss | | threatening |
| Symptoms-Other (Specify, Alopecia Bruising (in absence of grade 3 or 4 thrombocytopenia) | normal<br>none | DERMATOL mild hair loss localized or in dependent area | OGY/SKIN pronounced hair loss | - | threatening<br>or disabling<br>- |

| | | Grade | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2<br>moderate to brisk | 3<br>confluent moist | 4<br>skin |
| Dermatitis, focal (associated with high-dose chemotherapy and bone marrow transplant) | none | faint erythema or<br>dry<br>desquamation | erythema or a patchy moist desquamation, mostly confined to skin folds and creases; moderate edema | desquamation, ≥1.5 cm diameter, not confined to skin folds; pitting edema | necrosis or<br>ulceration of<br>full<br>thickness<br>dermis; may<br>include<br>spontaneou<br>s bleeding<br>not induced<br>by minor<br>trauma or<br>abrasion |
| Dry skin | normal | controlled with emollients | not controlled<br>with emollients | - | - |
| Erythema<br>multiforme (e.g.,<br>Stevens-Johnson<br>syndrome, toxic<br>epidermal<br>necrolysis) | absent | - | scattered, but not<br>generalized<br>eruption | severe or<br>requiring IV<br>fluids (e.g.,<br>generalized rash<br>or painful<br>stomatitis) | life-<br>threatening<br>(e.g.,<br>exfoliative<br>or<br>ulcerating<br>dermatitis<br>or requiring<br>enteral or<br>parenteral<br>nutritional<br>support) |
| Flushing | absent | present | - | - | - |
| Hand-foot skin<br>reaction | none | skin changes or<br>dermatitis<br>without pain<br>(e.g., erythema,<br>peeling) | skin changes<br>with pain, not<br>interfering with<br>function | skin changes<br>with pain,<br>interfering with<br>function | - |
| Injection site reaction | none | pain or itching or<br>erythema | pain or swelling,<br>with<br>inflammation or<br>phlebitis | ulceration or<br>necrosis that is<br>severe or<br>prolonged, or<br>requiring surgery | - |
| Nail changes | normal | discoloration or<br>ridging<br>(koilonychia) or<br>pitting | partial or<br>complete loss of<br>nail(s) or pain in<br>nailbeds | _ | • |
| Petechiae is graded i | n the HEMORR | | | | |
| Photosensitivity | none | painless<br>erythema | painful erythema | erythema with desquamation | - |
| Pigmentation<br>changes (e.g.,<br>vitiligo) | none | localized<br>pigmentation<br>changes | generalized<br>pigmentation<br>changes | - | - |
| Pruritus Purpura is graded in | none | mild or localized, relieved spontaneously or by local measures | intense or<br>widespread,<br>relieved<br>spontaneously or<br>by systemic<br>measures | intense or<br>widespread and<br>poorly controlled<br>despite treatment | - |

| | | Grad | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Radiation dermatitis Note: Pain associated | none | faint erythema or<br>dry<br>desquamation | moderate to brisk erythema or a patchy moist desquamation, mostly confined to skin folds and creases; moderate edema | confluent moist desquamation, ≥1.5 cm diameter, not confined to skin folds; pitting edema | skin necrosis or ulceration o full thickness dermis; may include bleeding no induced by minor trauma or abrasion |
| radiation. | Willi Tadiation GC | matrib io graded bej | paratery in the 171111 | category as runi aut | . 10 |
| Radiation recall reaction (reaction following chemotherapy in the absence of additional radiation therapy that occurs in a previous radiation port) | none | faint erythema or<br>dry<br>desquamation | moderate to brisk<br>erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases;<br>moderate edema | confluent moist<br>desquamation,<br>≥1.5 cm diameter,<br>not confined to<br>skin folds; pitting<br>edema | skin necrosis or ulceration of full thickness dermis; may include bleeding not induced by minor trauma or abrasion |
| Rash/desquamation | none | macular or papular eruption or erythema without associated symptoms | macular or papular eruption or erythema with pruritus or other associated symptoms covering <50% of body surface or localized desquamation or other lesions covering <50% of body surface area | symptomatic<br>generalized<br>erythroderma or<br>macular, papular<br>or vesicular<br>eruption or<br>desquamation<br>covering ≥50% of<br>body surface area | generalized<br>exfoliative<br>dermatitis<br>or ulcerative<br>dermatitis |
| For BMT: | none | macular or<br>papular eruption<br>or erythema<br>covering <25% of<br>body surface area<br>without<br>associated<br>symptoms | macular or papular eruption or erythema with pruritis or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area | symptomatic generalized erythroderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering ≥50% of body surface area | generalized<br>exfoliative<br>dermatitis<br>or ulcerative<br>dermatitis<br>or bullous<br>formation |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Urticaria<br>(hives, welts,<br>wheals) | none | requiring no<br>medication | requiring PO or<br>topical treatment<br>or IV medication<br>or steroids for<br><24 hours | requiring IV<br>medication or<br>steroids for ≥24<br>hours | - |
| Wound- infectious | none | cellulitis | superficial<br>infection | infection<br>requiring IV<br>antibiotics | necrotizing<br>fascitis |
| Wound- non-<br>infectious | none | incisional<br>separation | incisional hernia | fascial disruption<br>without<br>evisceration | fascial<br>disruption<br>with<br>evisceration |
| Dermatology/Skin-<br>Other<br>(Specify,) | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | ENDOCI | RINE | | |
| Cushingoid appearance (e.g., moon face with or without buffalo hump, centripetal obesity, cutaneous | absent | - | present | | • |
| striae)<br>Also consider Hyperg | lycemia, Hypoka | lemia. | | | |
| Feminization of male | absent | - | - | present | |
| Gynecomastia | none | mild | pronounced or<br>painful | pronounced or<br>painful and<br>requiring surgery | - |
| Hot flashes/flushes | none | mild or no more<br>than 1 per day | moderate and<br>greater than 1 per<br>day | - | - |
| Hypothyroidism | absent | asymptomatic,TS<br>H elevated, no<br>therapy given | symptomatic or<br>thyroid<br>replacement<br>treatment given | patient<br>hospitalized for<br>manifestations of<br>hypothyroidism | myxedema<br>coma |
| Masculinization of female | absent | - | - | present | - |
| SIADH (syndrome<br>of inappropriate<br>antidiuretic<br>hormone) | absent | - | - | present | • |
| Endocrine-Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | GASTROINT | | | |
| Amylase is graded in | the METABOLIC | | egory. | | |
| Anorexia | none | loss of appetite | oral intake<br>significantly<br>decreased | requiring IV<br>fluids | requiring<br>feeding tube<br>or<br>parenteral<br>nutrition |

| Toxicity | | Grad | C | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Ascites (non-<br>malignant) | none | asymptomatic | symptomatic,<br>requiring<br>diuretics | symptomatic,<br>requiring<br>therapeutic<br>paracentesis | life-<br>threatening<br>physiologic<br>consequenc |
| Colitis | nono | | ahdominal nain | ahdominal nain | es |
| | none | | abdominal pain<br>with mucus<br>and/or blood in<br>stool | abdominal pain,<br>fever, change in<br>bowel habits<br>with ileus or<br>peritoneal signs,<br>and radiographic<br>or biopsy<br>documentation | perforation<br>or requiring<br>surgery or<br>toxic<br>megacolon |
| | | ng with grade 3 or 4 throi | | | thout grade |
| 3 or 4 infombocytope<br>Constipation | none | GI bleeding, Rectal bleedi<br>requiring stool | requiring | obstipation | obstruction |
| Consupation | HOHE | softener or | laxatives | requiring manual | or toxic |
| | a constant | dietary - | ianaii v Co | evacuation or | megacolon |
| | | modification | | enema | 1110001021 |
| Dehydration | none | dry mucous | requiring IV fluid | requiring IV fluid | physiologic |
| | 1010 | membranes<br>and/or<br>diminished skin<br>turgor | replacement<br>(brief) | replacement<br>(sustained) | consequences requiring intensive care; hemodyna |
| 4.1 .1 TYDOU . | . 5. 1 | 77 ''' × 0' ''' | /oc1 | 20.000000 1 1.1 V | mic collapse |
| | | ea, Vomiting, Stomatitis, | | | • |
| Diarrhea<br>Patients without | ension, Diarrho<br>none | ea, Vomiting, Stomatitis,<br>increase of < 4<br>stools/day over<br>pre-treatment | pharyngitis (oral/pl<br>increase of 4-6<br>stools/day, or<br>nocturnal stools | increase of ≥7 stools/day or incontinence; or need for parenteral support for | physiologic<br>consequenc<br>es requiring<br>intensive<br>care; or<br>hemodyna |
| Diarrhea Patients without colostomy: Patients with a | | increase of < 4<br>stools/day over | increase of 4-6 stools/day, or nocturnal stools moderate increase in loose, watery colostomy output compared with pretreatment, but not interfering with normal | increase of ≥7<br>stools/day or<br>incontinence; or<br>need for<br>parenteral | physiologic<br>consequence<br>es requiring<br>intensive<br>care; or<br>hemodyna<br>mic collapse<br>physiologic<br>consequence<br>es, requiring<br>intensive<br>care; or<br>hemodyna |
| Also consider Hypot Diarrhea Patients without colostomy: Patients with a colostomy: | none | increase of < 4 stools/day over pre-treatment mild increase in loose, watery colostomy output compared with | increase of 4-6 stools/day, or nocturnal stools moderate increase in loose, watery colostomy output compared with pretreatment, but not interfering | increase of ≥7 stools/day or incontinence; or need for parenteral support for dehydration severe increase in loose, watery colostomy output compared with pretreatment, interfering with | physiologic<br>consequence<br>es requiring<br>intensive<br>care; or<br>hemodyna<br>mic collapse<br>physiologic<br>consequence<br>es, requiring<br>intensive<br>care; or |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Duodenal ulcer<br>(requires<br>radiographic or<br>endoscopic<br>documentation) | none | _ | requiring<br>medical<br>management or<br>non-surgical<br>treatment | uncontrolled by outpatient medical management; requiring hospitalization | perforation<br>or bleeding,<br>requiring<br>emergency<br>surgery |
| Dyspepsia/heartbur<br>n | none | mild | moderate | severe | - |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If toxicity is rad | none | mild dysphagia,<br>but can eat<br>regular diet<br>grade <u>either</u> under Dys | dysphagia, requiring predominantly pureed, soft, or liquid diet sphagia- esophageal r | dysphagia,<br>requiring IV<br>hydration<br>related to radiation <u>or</u> | complete obstruction (cannot swallow saliva) requiring enteral or parenteral nutritional support, or perforation Dysphagia- |
| pharyngeal related to | radiation. | | | | |
| Dysphagia- esophageal related to radiation Also consider Pain du | none | mild dysphagia, but can eat regular diet Mucositis due to radia | dysphagia, requiring predominantly liquid, pureed or soft diet | dysphagia<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Note: Fistula is grade | | | | | |
| Dysphagia - pharyngeal related to radiation Also consider Pain du | none | mild dysphagia, but can eat regular diet Mucositis due to radia | dysphagia, requiring predominantly pureed, soft, or liquid diet | dysphagia,<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Note: Fistula is grade | d separately as | | PACA M | nrocent | noguiein a |
| Fistula- esophageal | none | | <u>-</u> | present | requiring<br>surgery |
| Fistula- intestinal | | | _ | | requiring |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Fistula- pharyngeal | none | - | - | present | requiring<br>surgery |
| Fistula- rectal/anal | none | - | - | present | requiring<br>surgery |
| Flatulence | none | mild | moderate | - | - |
| Gastric ulcer<br>(requires<br>radiographic or<br>endoscopic<br>documentation) | none | - | requiring<br>medical<br>management or<br>non-surgical<br>treatment | bleeding without perforation, uncontrolled by outpatient medical management; requiring hospitalization or | perforation<br>or bleeding,<br>requiring<br>emergency<br>surgery |
| Also consider Hemor<br>3 or 4 thrombocytope | | vith grade 3 or 4 thro | mbocytopenia, Hemo | surgery<br>orrhage/bleeding wi | thout grade |
| Gastritis | none | - | requiring<br>medical<br>management or<br>non-surgical<br>treatment | uncontrolled by out-patient medical management; requiring hospitalization or surgery | life-<br>threatening<br>bleeding,<br>requiring<br>emergency<br>surgery |
| Also consider Hemor<br>3 or 4 thrombocytope<br>Hematemesis is grad<br>Hematochezia is grad | nia.<br>ed in the HEMOR | RHAGE category. | | | |
| Ileus (or<br>neuroconstipation) | none | - | intermittent, not requiring intervention | requiring non-<br>surgical<br>intervention | requiring<br>surgery |
| Mouth dryness | normal | mild | moderate | • | - |
| Esophagitis, Gas<br>RENAL/GENII | stritis, Stomatitis,<br>OURINARY cate | is graded in the GAS<br>pharyngitis (oral/ph<br>gory for Vaginititis,<br>ided as Mucositis due<br>erythema of the<br>mucosa | patchy<br>pseudomembran | ategory for specific si<br>and Typhlitis; or the<br>confluent<br>pseudomembran<br>ous reaction | necrosis or deep |
| | | | ous reaction<br>(patches<br>generally ≤ 1.5<br>cm in diameter<br>and non-<br>contiguous) | (contiguous patches generally > 1.5 cm in diameter) | ulceration;<br>may include<br>bleeding no<br>induced by<br>minor<br>trauma or |
| Dysphagia relat | ion mucositis of t<br>ed to radiation is | also graded as either | (patches<br>generally ≤ 1.5<br>cm in diameter<br>and non- | (contiguous patches generally > 1.5 cm in diameter) | ulceration;<br>may include<br>bleeding not<br>induced by<br>minor<br>trauma or<br>abrasion |

| | | Grade | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Pancreatitis | none | - | - | abdominal pain<br>with pancreatic<br>enzyme elevation | complicated<br>by shock<br>(acute<br>circulatory<br>failure) |
| Also consider Hypoter<br>Note: Asymptomatic a | mylase and Amy | lase are graded in th | e METABOLIC/LAE | ORATORY category | <u> </u> |
| Pharyngitis is graded i<br>mucositis). | n the GASTROIN | NTESTINAL category | | ngitis (oral/pharynខ្ | geal |
| Proctitis | none | increased stool frequency, occasional blood- streaked stools, or rectal discomfort (including hemorrhoids), not requiring medication | increased stool<br>frequency,<br>bleeding, mucus<br>discharge, or<br>rectal discomfort<br>requiring<br>medication; anal<br>fissure | increased stool frequency/diarrh ea, requiring parenteral support; rectal bleeding, requiring transfusion; or persistent mucus discharge, necessitating pads | perforation,<br>bleeding or<br>necrosis or<br>other life-<br>threatening<br>complication<br>n requiring<br>surgical<br>intervention<br>(e.g.,<br>colostomy) |
| Proctitis occurrin<br>Late Radiation M<br>Salivary gland | iia, and Pain due<br>ed separately as :<br>g more than 90 d | to radiation. Fistula- rectal/anal. ays after the start of Scheme. (See Appen slightly | radiation therapy is &dix IV) thick, ropy, | | /EORTC |
| changes | | thickened saliva/may have slightly altered taste (e.g., metallic); additional fluids may be required | sticky saliva;<br>markedly altered<br>taste; alteration<br>in diet required | | salivary<br>gland<br>necrosis |
| Sense of smell | normal | slightly altered | markedly altered | - | - |
| Stomatitis/pharyngi<br>tis (oral/pharyngeal<br>mucositis) | none | painless ulcers,<br>erythema, or<br>mild soreness in<br>the absence of<br>lesions | painful erythema, edema, or ulcers, but can eat or swallow | painful<br>erythema,<br>edema, or ulcers<br>requiring IV<br>hydration | severe ulceration or requires parenteral or enteral nutritional support or prophylatic intubation |
| For BMT: | none | painless ulcers,<br>erythema, or<br>mild soreness in<br>the absence of<br>lesions | painful<br>erythema, edema<br>or ulcers but can<br>swallow | painful erythema, edema, or ulcers preventing swallowing or requiring hydration or parenteral (or enteral) nutritional support | severe ulceration requiring prophylactic intubation or resulting in documented aspiration pneumonia |

| | | Grade | 9 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: Radiation-related | d mucositis is gra | ded as Mucositis due | e to radiation. | | |
| Taste disturbance (dysgeusia) | normal | slightly altered | markedly altered | - | - |
| Typhlitis (inflammation of the cecum) | none | - | - | abdominal pain,<br>diarrhea, fever,<br>or radiographic<br>documentation | perforation,<br>bleeding or<br>necrosis or<br>other life-<br>threatening<br>complicatio<br>n requiring<br>surgical<br>intervention<br>(e.g.,<br>colostomy) |
| Also consider Hemorr<br>3 or 4 thrombocytoper | hage/bleeding w<br>iia, Hypotension, | ith grade 3 or 4 throi<br>Febrile/neutropenia | i. | | |
| Vomiting Also consider Dehydr | none | 1 episode in 24<br>hours over<br>pretreatment | 2-5 episodes in 24<br>hours over<br>pretreatment | ≥6 episodes in 24 hours over pretreatment; or need for IV fluids | Requiring parenteral nutrition; or physiologic consequenc es requiring intensive care; hemodyna mic collapse |
| Weight gain is graded | in the CONSTIT | UTIONAL SYMPTO | MS category. | | |
| Weight loss is graded | in the CONSTITU | | | | *** |
| Gastrointestinal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | HEMORR | HAGE | | |
| For <u>any</u> bleeding 4 thrombocytope grade that incorp If the site or type bleeding: CNS he surgery, Melena, bleeding/hemate If the platelet cou | with grade 3 or 4 cmia. Also consider or a consider of hemorrhage/lemorrhage/lemorrhage/lower GI bleedir ochezia, Vaginal lant is ≥50,000 and and the platelet of | r platelets, transfusion type of bleeding. bleeding is listed, alsoling, Hematuria, Hemag, Petechiae/purpurbleeding. the site or type of bleeding is the site or type of bleeding. | always grade Hemonon-pRBCS, and transformers of use the grading that the grading that the grading is Hemoptys of the grading is listed, grading is listed, grading Hemorrhage/bleed THER category. | fusion-platelets in act<br>it incorporates the sit<br>sis, Hemorrhage/ble<br>eding into skin), Rect<br>e the specific site. If | Idition to the te of eding with al the site or |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hemorrhage/bleedi<br>ng with grade 3 or 4<br>thrombocytopenia | none | mild without<br>transfusion | | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Note: This toxicity m | nust be graded | Transfusion-platelet, T<br>for any bleeding with §<br>f the site is not listed, g | grade 3 or 4 thromb | ocytopenia. Also grad<br>HEMORRHAGE cate | e the site or |
| Hemorrhage/bleedi<br>ng without grade 3<br>or 4<br>thrombocytopenia | none | mild without<br>transfusion | | requiring<br>transfusion | catastrophic<br>bleeding<br>requiring<br>major non-<br>elective<br>intervention |
| Note: Bleeding in th | e absence of gr<br>sted elsewhere | Transfusion-platelet, Tade 3 or 4 thrombocyto in the HEMORRHAGE | penia is graded her | e only if the specific s<br>de as Other in the | |
| CNS<br>hemorrhage/bleedin<br>g | none | - | - | bleeding noted<br>on CT or other<br>scan with no<br>clinical<br>consequences | hemorrhagi<br>c stroke or<br>hemorrhagi<br>c vascular<br>event (CVA)<br>with<br>neurologic<br>signs and<br>symptoms |
| Epistaxis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematemesis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematuria<br>(in the absence of<br>vaginal bleeding) | none | microscopic only | intermittent<br>gross bleeding,<br>no clots | persistent gross<br>bleeding or clots;<br>may require<br>catheterization or<br>instrumentation,<br>or transfusion | open<br>surgery or<br>necrosis or<br>deep<br>bladder<br>ulceration |
| Hemoptysis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hemorrhage/bleeding associated with surgery Note: Expected blood | none | mild without<br>transfusion | d as a toxicity. | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Melena/GI bleeding | none | mild without | - | requiring | catastrophic |
| wielena/ Grotecung | none | transfusion | | transfusion | bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Petechiae/purpura<br>(hemorrhage/bleedi<br>ng into skin or<br>mucosa) | none | rare petechiae of<br>skin | petechiae or<br>purpura in<br>dependent areas<br>of skin | generalized petechiae or purpura of skin or petechiae of any mucosal site | - |
| Rectal bleeding/<br>hematochezia | none | mild without<br>transfusion or<br>medication | persistent, requiring medication (e.g., steroid suppositories) and/or break from radiation treatment | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Vaginal bleeding | none | spotting,<br>requiring < 2<br>pads per day | requiring ≥ 2<br>pads per day, but<br>not requiring<br>transfusion | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hemorrhage-Other<br>(Specify site,<br>) | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| | | HEPAT | TC | | |
| Alkaline<br>phosphatase | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5.0 x ULN | > 5.0 - 20.0 x<br>ULN | > 20.0 x<br>ULN |
| Bilirubin | WNL | > ULN - 1.5 x<br>ULN | > 1.5 - 3.0 x ULN | > 3.0 - 10.0 x<br>ULN | > 10.0 x<br>ULN |
| Bilirubin- graft versus | | HD) | | | |
| Note: The following cr | riteria are used on<br>normal | lly for bilirubin assoc<br>≥2 - <3 mg/100<br>ml | iated with graft vers<br>≥3 - <6 mg/100<br>ml | us host disease.<br>≥6 - <15 mg/100<br>ml | ≥15 mg/100<br>ml |
| GGT<br>(γ - Glutamyl<br>transpeptidase) | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5.0 × ULN | > 5.0 - 20.0 x<br>ULN | > 20.0 x<br>ULN |
| Hepatic enlargement<br>Note: Grade Hepatic e | absent<br>nlargement only | -<br>for changes related to | o VOD or other treat | present<br>ment related toxicity. | - |
| Tiotel Orage Trefatte c | | | ≥2 - <3 g/dl | | |

| | | Grad | ic | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | _ 2 | 3 | 4 |
| Liver<br>dysfunction/failure<br>(clinical) | normal | - I I I I I I I I I I I I I I I I I I I | ON salasass | asterixis | encephalopa<br>thy or coma |
| | | graded in the INFECTI | ON category. | | |
| Portal vein flow | normal | - | decreased portal<br>vein flow | reversal/retrogra<br>de portal vein<br>flow | - |
| SGOT (AST)<br>(serum glutamic<br>oxaloacetic<br>transaminase) | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5.0 x ULN | > 5.0 - 20.0 x<br>ULN | > 20.0 x<br>ULN |
| SGPT (ALT)<br>(serum glutamic<br>pyruvic<br>transaminase) | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5.0 x ULN | > 5.0 - 20.0 x<br>ULN | > 20.0 x<br>ULN |
| Hepatic-Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| <del></del> | | INFECTION/FEBRIL | E NEUTROPENIA | | |
| Catheter-related infection | none | mild, no active<br>treatment | moderate, localized infection, requiring local or oral treatment | severe, systemic infection, requiring IV antibiotic or antifungal treatment or hospitalization | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection) (ANC < 1.0 x 10 <sup>9</sup> /L, fever ≥38.5°C) | none | may be associated with | neutropenia and is | Present | Life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| | | may be associated with | Theutroperua and 15 g | | life- |
| Infection<br>(documented<br>clinically or<br>microbiologically)<br>with grade 3 or 4 | none | - | - | present | threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| neutropenia<br>(ANC < 1.0 x 10 <sup>9</sup> /L)<br>Note: Hypothermia<br>documented infe | instead of fevection with gra | er may be associated w<br>ide 3 or 4 neutropenia, | rith neutropenia and i<br>grade as Febrile neutr | s graded here. In the<br>openia. | absence of |
| Infection with<br>unknown ANC | none<br>terion is used | - | - | present | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Infection without neutropenia | none | mild, no active<br>treatment | moderate,<br>localized<br>infection,<br>requiring local or<br>oral treatment | severe, systemic infection, requiring IV antibiotic or antifungal treatment, or hospitalization | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| Infection/Febrile<br>Neutropenia-Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| Wound-infectious is gr | aded in the DER | MATOLOGY/SKIN | category. | | |
| | | LYMPHA | TICS | | |
| Lymphatics | normal | mild<br>lymphedema | moderate<br>lymphedema<br>requiring<br>compression;<br>lymphocyst | severe<br>lymphedema<br>limiting function;<br>lymphocyst<br>requiring surgery | severe lymphedem a limiting function with ulceration |
| Lymphatics-Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | METABOLIC/LA | BORATORY | | |
| Acidosis<br>(metabolic or<br>respiratory) | normal | pH < normal, but<br>≥7.3 | - | pH < 7.3 | pH < 7.3<br>with life-<br>threatening<br>physiologic<br>consequenc<br>es |
| Alkalosis<br>(metabolic or<br>respiratory) | normal | pH > normal, but<br>≤7.5 | - | pH > 7.5 | pH > 7.5<br>with life-<br>threatening<br>physiologic<br>consequenc<br>es |
| Amylase | WNL | > ULN - 1.5 x<br>ULN | > 1.5 - 2.0 x ULN | > 2.0 - 5.0 x ULN | >5.0 x ULN |
| Bicarbonate | WNL | < LLN - 16<br>mEq/dl | 11 - 15 mEq/dl | 8 - 10 mEq/dl | < 8 mEq/dl |
| CPK<br>(creatine<br>phosphokinase) | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5 x ULN | > 5 - 10 x ULN | > 10 x ULN |
| Hypercalcemia | WNL | > ULN - 11.5<br>mg/dl<br>> ULN - 2.9<br>mmol/L | >11.5 - 12.5<br>mg/dl<br>> 2.9 - 3.1<br>mmol/L | >12.5 - 13.5<br>mg/dl<br>> 3.1 - 3.4<br>mmol/L | > 13.5<br>mg/dl<br>> 3.4<br>mmol/L |
| Hypercholesterolemi<br>a | WNL | > ULN - 300<br>mg/dl<br>> ULN - 7.75<br>mmol/L | > 300 - 400<br>mg/dl<br>> 7.75 - 10.34<br>mmol/L | > 400 - 500<br>mg/dl<br>>10.34 - 12.92<br>mmol/L | > 500 mg/dl<br>> 12.92<br>mmol/L |
| Hyperglycemia | WNL | > ULN - 160<br>mg/dl<br>> ULN - 8.9<br>mmol/L | > 160 - 250<br>mg/dl<br>> 8.9 - 13.9<br>mmol/L | > 250 - 500<br>mg/dl<br>> 13.9 - 27.8<br>mmol/L | > 500 mg/dl<br>> 27.8<br>mmol/L or<br>ketoacidosis |

| | | Grade | 2 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hyperkalemia | WNL | > ULN - 5.5 | > 5.5 - 6.0 | > 6.0 - 7.0 | > 7.0 |
| 71 | | mmol/L | mmol/L | mmol/L | mmol/L |
| Hypermagnesemia | WNL | > ULN - 3.0 | - | $> 3.0 - 8.0 \mathrm{mg/dl}$ | > 8.0 mg/dl |
| 71 0 | | mg/dl | | > 1.23 - 3.30 | > 3.30 |
| | | > ULN - 1.23 | | mmol/L | mmol/L |
| | | mmol/L | | | |
| Hypernatremia | WNL | > ULN - 150 | >150 - 155 | >155 - 160 | >160 |
| | | mmol/L | mmol/L | mmol/L | mmol/L |
| Hypertriglyceridemi<br>a | WNL | > ULN - 2.5 x<br>ULN | > 2.5 - 5.0 x ULN | > 5.0 - 10 x ULN | > 10 x ULN |
| Hyperuricemia | WNL | > ULN - ≤ 10 | - | > ULN - ≤ 10 | > 10 mg/dl |
| | | mg/dl | | mg/dl | > 0.59 |
| | | $\leq 0.59 \text{mmol/L}$ | | $\leq 0.59 \text{ mmol/L}$ | mmol/L |
| | | without | | with physiologic | |
| | | physiologic | | consequences | |
| | | consequences | | | |
| Also consider Tumor l | ysis syndrome, I | Renal failure, Creatini | ne, Potassium. | | |
| Hypocalcemia | WNL | <lln -="" 8.0<="" td=""><td>7.0 - &lt; 8.0 mg/dl</td><td>6.0 - &lt; 7.0 mg/dl</td><td>&lt;6.0 mg/dl</td></lln> | 7.0 - < 8.0 mg/dl | 6.0 - < 7.0 mg/dl | <6.0 mg/dl |
| | | mg/dl | 1.75 - < 2.0 | 1.5 - < 1.75 | < 1.5 |
| | | <lln -="" 2.0<="" td=""><td>mmol/L</td><td>mmol/L</td><td>mmol/L</td></lln> | mmol/L | mmol/L | mmol/L |
| | | mmol/L | | | |
| Hypoglycemia | WNL | <lln -="" 55="" dl<="" mg="" td=""><td>40 - &lt; 55 mg/dl</td><td>30 - &lt; 40 mg/dl</td><td>&lt; 30 mg/dl</td></lln> | 40 - < 55 mg/dl | 30 - < 40 mg/dl | < 30 mg/dl |
| | | <lln -="" 3.0<="" td=""><td>2.2 - &lt; 3.0</td><td>1.7 - &lt; 2.2</td><td>&lt; 1.7</td></lln> | 2.2 - < 3.0 | 1.7 - < 2.2 | < 1.7 |
| | | mmol/L | mmol/L | mmol/L | mmol/L |
| Hypokalemia | WNL | <lln -="" 3.0<="" td=""><td>~</td><td>2.5 - &lt;3.0</td><td>&lt;2.5</td></lln> | ~ | 2.5 - <3.0 | <2.5 |
| | | mmol/L | 00 10 /11 | mmol/L | mmol/L |
| Hypomagnesemia | WNL | <lln -="" 1.2<="" td=""><td>0.9 - &lt;1.2 mg/dl</td><td>0.7 - &lt; 0.9 mg/dl</td><td>&lt; 0.7 mg/dl</td></lln> | 0.9 - <1.2 mg/dl | 0.7 - < 0.9 mg/dl | < 0.7 mg/dl |
| | | mg/dl | 0.4 - < 0.5 | 0.3 - < 0.4 | < 0.3 |
| | | <lln -="" 0.5<="" td=""><td>mmol/L</td><td>mmol/L</td><td>mmol/L</td></lln> | mmol/L | mmol/L | mmol/L |
| ** | XATA II | mmol/L | | 120 - <130 | <120 |
| Hyponatremia | WNL | <lln -="" 130<="" td=""><td>-</td><td>mmol/L</td><td>mmol/L</td></lln> | - | mmol/L | mmol/L |
| TT 1 1 ( ' | TATE IT | mmol/L | >20 <25 ma/dl | ≥1.0 - <2.0 mg/dl | < 1.0 mg/dl |
| Hypophosphatemia | WNL | <lln -2.5="" dl<="" mg="" td=""><td>≥2.0 - &lt;2.5 mg/d1<br/>≥0.6 - &lt;0.8</td><td>≥1.0 - &lt;2.0 mg/ ai<br/>≥0.3 - &lt;0.6</td><td>&lt; 1.0 Hig/ til</td></lln> | ≥2.0 - <2.5 mg/d1<br>≥0.6 - <0.8 | ≥1.0 - <2.0 mg/ ai<br>≥0.3 - <0.6 | < 1.0 Hig/ til |
| | | <lln -="" 0.8<="" td=""><td>≥0.6 - &lt;0.8<br/>mmol/L</td><td></td><td>mmol/L</td></lln> | ≥0.6 - <0.8<br>mmol/L | | mmol/L |
| TT .1 .1. | 1 1: (1 TATE) | mmol/L | mmoi/L | mmol/L | HIIIOI/L |
| Hypothyroidism is gra | | OCKINE category. | > 1.5 - 2.0 x ULN | > 2.0 - 5.0 x ULN | > 5.0 x ULN |
| Lipase | WNL | > ULN - 1.5 x<br>ULN | | > 2.0 - 5.0 X ULIN | |
| Metabolic/Laborator | none | mild | moderate | severe | life- |
| y-Other (Specify, | | | | | threatening |
| | | | | | or disabling |
| | | MUSCULOSI | KELETAL | | |
| Arthralgia is graded in | | | 1 | | 11 1.11 |
| Arthritis | none | mild pain with | moderate pain | severe pain with | disabling |
| | | inflammation, | with | inflammation, | |
| | | erythema or joint | inflammation, | erythema, or | |
| | | swelling but not | erythema, or | joint swelling | |
| | | interfering with | joint swelling | and interfering | |
| | | function | interfering with | with activities of | |
| | | | function, but not | daily living | |
| | | | interfering with<br>activities of daily | | |
| | | | living | | |
| | | | nvmg | | |

| | | Grad | e a | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Muscle weakness<br>(not due to<br>neuropathy) | normal | asymptomatic<br>with weakness<br>on physical exam | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | bedridden<br>or disabling |
| Myalgia is graded in t | he PAIN category | | | | |
| Myositis<br>(inflammation/dam<br>age of muscle) | none | mild pain, not interfering with function | pain interfering with function, but not interfering with activities of daily living | pain interfering<br>with function<br>and interfering<br>with activities of<br>daily living | bedridden<br>or disabling |
| Also consider CPK. | 1 1 55 | /: 1 / 1 CDY/ | | | |
| Note: Myositis implies | | | armatanatic ar 1 | armantamatic ar i | armantamati |
| Osteonecrosis<br>(avascular necrosis) | none | asymptomatic<br>and detected by<br>imaging only | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | symptomati<br>c; or<br>disabling |
| Musculoskeletal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | NEUROL | | | |
| Aphasia, receptive and | d/or expressive, i | s graded under Spee | ch impairment in the | | gory. |
| Arachnoiditis/meni<br>ngismus/<br>radiculitis | absent | mild pain not interfering with function | moderate pain interfering with function, but not interfering with activities of daily living | severe pain<br>interfering with<br>activities of daily<br>living | unable to<br>function or<br>perform<br>activities of<br>daily living;<br>bedridden;<br>paraplegia |
| Also consider Headac | he, Vomiting, Fev | | | | |
| Ataxia<br>(incoordination) | normal | asymptomatic<br>but abnormal on<br>physical exam,<br>and not<br>interfering with<br>function | mild symptoms interfering with function, but not interfering with activities of daily living | moderate<br>symptoms<br>interfering with<br>activities of daily<br>living | bedridden<br>or disabling |
| CNS cerebrovascular ischemia | none | - | - | transient<br>ischemic event or<br>attack (TIA) | permanent<br>event (e.g.,<br>cerebral<br>vascular<br>accident) |
| CNS hemorrhage/ble | eding is graded i | n the HEMORRHAG | E category. | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Cognitive disturbance/<br>learning problems | none | cognitive disability; not interfering with work/school performance; preservation of intelligence | cognitive disability; interfering with work/school performance; decline of 1 SD (Standard Deviation) or loss of developmental | cognitive disability; resulting in significant impairment of work/school performance; cognitive decline > 2 SD | inability to<br>work/frank<br>mental<br>retardation |
| Confusion | normal | confusion or | milestones<br>confusion or | confusion or | harmful to |
| Contusion | HOIMAI | disorientation or<br>attention deficit<br>of brief duration;<br>resolves<br>spontaneously<br>with no sequelae | disorientation or<br>attention deficit<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | delirium<br>interfering with<br>activities of daily<br>living | others or<br>self;<br>requiring<br>hospitalizat |
| Cranial neuropathy is | graded in the NE | UROLOGY category | | ial. | |
| Delusions | normal | _ | - | present | toxic<br>psychosis |
| Depressed level of consciousness | normal | somnolence or<br>sedation not<br>interfering with<br>function | somnolence or<br>sedation<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | obtundation or<br>stupor; difficult<br>to arouse;<br>interfering with<br>activities of daily<br>living | coma |
| Note: Syncope (faintir | ng) is graded in the | | gory. | | |
| Dizziness/lighthead edness | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden<br>or disabling |
| Dysphasia, receptive a | and/or expressive | , is graded under Spe | | he NEUROLOGY ca | tegory. |
| Extrapyramidal/ involuntary movement/ restlessness | none | mild involuntary<br>movements not<br>interfering with<br>function | moderate involuntary movements interfering with function, but not interfering with activities of daily living | severe involuntary movements or torticollis interfering with activities of daily living | bedridden<br>or disabling |
| Hallucinations | normal | - | - | present | toxic<br>psychosis |
| Headache is graded ir<br>Insomnia | the PAIN categor<br>normal | ry.<br>occasional | difficulty | frequent | - |
| | | difficulty<br>sleeping not<br>interfering with<br>function | sleeping<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | difficulty<br>sleeping,<br>interfering with<br>activities of daily<br>living | |

| | | Grade | 2 | rage | |
|---|---|---|---|---|---|
| Taniaiku | 0 | 1 | 2 | a | 4 |
| Toxicity Irritability (children <3 years of age) | normal | mild; easily<br>consolable | moderate;<br>requiring<br>increased<br>attention | severe;<br>inconsolable | |
| Leukoencephalopathy<br>associated radiological<br>findings | normal | mild increase in SAS (subarachnoid space) and/or mild ventriculomegaly; and/or small (+/- multiple) focal T2 hyperintensities, involving periventricular white matter or < 1/3 of susceptible areas of cerebrum | moderate increase in SAS; and/or moderate ventriculomegaly; and/or focal T2 hyperintensities extending into centrum ovale; or involving 1/3 to 2/3 of susceptible areas of cerebrum | severe increase in SAS; severe ventriculomegaly; near total white matter T2 hyperintensities or diffuse low attenuation (CT); focal white matter necrosis (cystic) | severe increase in SAS; severe ventriculome galy; diffuse low attenuation with calcification (CT); diffuse white matter necrosis (MRI) amnesia |
| Memory loss | normai | interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | amnesia |
| Mood alteration-<br>anxiety agitation | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal<br>ideation or<br>danger to<br>self |
| Mood alteration-<br>depression | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood alteration interfering with function, but not interfering with activities of daily living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal<br>ideation or<br>danger to<br>self |
| Mood alteration-<br>euphoria | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood alteration interfering with function, but not interfering with activities of daily living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | danger to<br>self |
| Neuropathic pain is gr<br>Neuropathy- cranial | raded in the PAIN<br>absent | category. | present, not<br>interfering with<br>activities of daily<br>living | present,<br>interfering with<br>activities of daily<br>living | life-<br>threatening,<br>disabling |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Neuropathy- motor | normal | subjective<br>weakness but no<br>objective findings | mild objective weakness interfering with function, but not interfering with activities of daily living | objective<br>weakness<br>interfering with<br>activities of daily<br>living | paralysis |
| Neuropathy-sensory | normal | loss of deep<br>tendon reflexes<br>or paresthesia<br>(including<br>tingling) but not<br>interfering with<br>function | objective sensory loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living | sensory loss or<br>paresthesia<br>interfering with<br>activities of daily<br>living | permanent<br>sensory loss<br>that<br>interferes<br>with<br>function |
| Nystagmus<br>Also consider Vision-d | absent<br>louble vision. | present | and the second s | in 25 feet and an amount oberly followers. | ~- |
| Personality/behavio | normal | change, but not<br>disruptive to<br>patient or family | disruptive to patient or family | disruptive to<br>patient and<br>family; requiring<br>mental health<br>intervention | harmful to<br>others or<br>self;<br>requiring<br>hospitalizati<br>on |
| Pyramidal tract dysfunction (e.g., ↑ tone, hyperreflexia, positive Babinski, ↓ fine motor coordination) | normal | asymptomatic<br>with abnormality<br>on physical<br>examination | symptomatic or<br>interfering with<br>function but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden<br>or disabling<br>paralysis |
| Seizure(s) | none | - | seizure(s) self-<br>limited and<br>consciousness is<br>preserved | seizure(s) in<br>which<br>consciousness is<br>altered | seizures of<br>any type<br>which are<br>prolonged,<br>repetitive,<br>or difficult<br>to control<br>(e.g., status<br>epilepticus,<br>intractable<br>epilepsy) |
| Speech impairment<br>(e.g., dysphasia or<br>aphasia) | normal | - | awareness of<br>receptive or<br>expressive<br>dysphasia, not | receptive or<br>expressive<br>dysphasia,<br>impairing ability | inability to<br>communicate |

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 . | 2 | 3 | 4 |
| Tremor | none | mild and brief or<br>intermittent but<br>not interfering<br>with function | moderate tremor<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe tremor<br>interfering with<br>activities of daily<br>living | - |
| Vertigo | none | not interfering<br>with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden<br>or disabling |
| Neurology-Other<br>(Specify,<br>) | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | OCULAR/\ | /ISUAL | | |
| Cataract | none | asymptomatic | symptomatic,<br>partial visual loss | symptomatic, visual loss requiring treatment or interfering with function | - |
| Conjunctivitis . | none | abnormal ophthalmologic changes, but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Dry eye | normal | mild, not<br>requiring<br>treatment | moderate or<br>requiring<br>artificial tears | _ | - |
| Glaucoma | none | increase in<br>intraocular<br>pressure but no<br>visual loss | increase in<br>intraocular<br>pressure with<br>retinal changes | visual<br>impairment | unilateral or<br>bilateral loss<br>of vision<br>(blindness) |
| Keratitis<br>(corneal<br>inflammation/<br>corneal ulceration) | none | abnormal ophthalmologic changes but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | unilateral or<br>bilateral loss<br>of vision<br>(blindness) |
| Tearing (watery<br>eyes) | none | mild: not<br>interfering with<br>function | moderate: interfering with function, but not interfering with activities of daily living | interfering with<br>activities of daily<br>living | - |

| | | | | Page | |
|---|---|---|---|---|---|
| | | Grad | е . | | |
| Toxicity | 0 | _1 | 2 | 3 | 4 |
| Vision- blurred<br>vision | normal | - , | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | • |
| Vision- double<br>vision (diplopia) | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | - |
| Vision- flashing<br>lights/floaters | normal | mild, not<br>interfering with<br>function | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | _ |
| Vision- night<br>blindness<br>(nyctalopia) | normal | abnormal electro-<br>retinography but<br>asymptomatic | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | _ |
| Vision- photophobia | normal | _ | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | _ |
| Ocular/Visual-Other<br>(Specify,<br>) | normal | mild | moderate | severe | unilateral or<br>bilateral loss<br>of vision<br>(blindness) |
| | | PAIN | I | | |
| Abdominal pain or cramping | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Arthritis (joint pain wi | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain or analgesics severely interfering with activities of daily living LOSKELETAL category | disabling |

| | | Grad | le | | - |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Bone pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Chest pain<br>(non-cardiac and<br>non-pleuritic) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dysmenorrhea | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dyspareunia | none | mild pain not interfering with function | moderate pain<br>interfering with<br>sexual activity | severe pain<br>preventing<br>sexual activity | - |
| Dysuria is graded in | the RENAL/C | GENITOURINARY categ | ory. | | |
| Earache (otalgia) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Headache | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| | | Grade | | 1 age 3 | |
|---|---|---|---|---|---|
| Translation | 0 | | 2 | 3 | 4 |
| Toxicity Hepatic pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Myalgia<br>(muscle pain) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Neuropathic pain<br>(e.g., jaw pain,<br>neurologic pain,<br>phantom limb pain,<br>post-infectious<br>neuralgia, or painful<br>neuropathies) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pain due to radiation | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pelvic pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pleuritic pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| | | Grad | e = | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Rectal or perirectal<br>pain (proctalgia) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Tumor pain<br>(onset or<br>exacerbation of<br>tumor pain due to<br>treatment) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Tumor flair is graded | in the SYNIDRON | Æ category | living | | |
| Pain-Other<br>(Specify, | none | mild | moderate | severe | disabling |
| | | PULMON | JARY | | |
| Adult Respiratory<br>Distress Syndrome<br>(ARDS) | absent | - | - | - | present |
| Apnea | none | - | - | present | requiring intubation |
| Carbon monoxide<br>diffusion capacity<br>(DL <sub>CO</sub> ) | ≥ 90% of<br>pretreatment<br>or normal<br>value | ≥75 - <90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of pretreatment or normal value | < 25% of<br>pretreatmen<br>t or normal<br>value |
| Cough | absent | mild, relieved by<br>non-prescription<br>medication | requiring<br>narcotic<br>antitussive | severe cough or coughing spasms, poorly controlled or unresponsive to treatment | - |
| Dyspnea<br>(shortness of breath) | normal | - | dyspnea on<br>exertion | dyspnea at<br>normal level of<br>activity | dyspnea at<br>rest or<br>requiring<br>ventilator<br>support |
| FEV <sub>1</sub> | ≥ 90% of<br>pretreatment<br>or normal<br>value | ≥75 - <90% of<br>pretreatment or<br>normal value | ≥50 - <75% of<br>pretreatment or<br>normal value | ≥25 - <50% of<br>pretreatment or<br>normal value | < 25% of<br>pretreatmer<br>t or normal<br>value |
| Hiccoughs (hiccups,<br>singultus) | none | mild, not<br>requiring<br>treatment | moderate,<br>requiring<br>treatment | severe,<br>prolonged, and<br>refractory to<br>treatment | - |

| | | Grad | | - | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Нурохіа | normal | | decreased O <sub>2</sub><br>saturation with<br>exercise | decreased O <sub>2</sub> saturation at rest, requiring supplemental oxygen | decreased O <sub>2</sub> saturation, requiring pressure support (CPAP) or assisted ventilation |
| Pleural effusion<br>(non-malignant) | none | asymptomatic<br>and not requiring<br>treatment | symptomatic,<br>requiring<br>diuretics | symptomatic,<br>requiring O <sub>2</sub> or<br>therapeutic<br>thoracentesis | life-<br>threatening<br>(e.g.,<br>requiring<br>intubation) |
| Pleuritic pain is grade | d in the PAIN | | | | |
| Pneumonitis/pulmo<br>nary infiltrates | none | radiographic<br>changes but<br>asymptomatic or<br>symptoms not<br>requiring<br>steroids | radiographic<br>changes and<br>requiring<br>steroids or<br>diuretics | radiographic<br>changes and<br>requiring oxygen | radiographi<br>c changes<br>and<br>requiring<br>assisted<br>ventilation |
| Pneumothorax | none | no intervention | chest tube | sclerosis or | life- |
| | | required | required | surgery required | threatening |
| | is graded as Tl | nrombosis/embolism ir | the CARDIOVASCI | | |
| Pulmonary fibrosis | none | radiographic<br>changes, but<br>asymptomatic or<br>symptoms not<br>requiring<br>steroids | requiring<br>steroids or<br>diuretics | requiring oxygen | requiring<br>assisted<br>ventilation |
| Note: Radiation-relate<br>Scheme- Lung. (See A | d pulmonary f<br>ppendix IV) | ibrosis is graded in the | | | |
| Voice<br>changes/stridor/lar<br>ynx (e.g., hoarseness,<br>loss of voice,<br>laryngitis) | normal | mild or<br>intermittent<br>hoarseness | persistent<br>hoarseness, but<br>able to vocalize;<br>may have mild to<br>moderate edema | whispered<br>speech, not able<br>to vocalize; may<br>have marked<br>edema | marked dyspnea/st idor requiring tracheostom y or intubation |
| Radiation-related | l hemoptysis fi<br>TNAL categor | ded as cough in the PUT<br>com larynx/pharynx is<br>y. Radiation-related he<br>HAGE category. | graded as Grade 4 M | lucositis due to radia | tion in the |
| Pulmonary-Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |

| | | | | Page | 00 |
|---|---|---|---|---|---|
| | | Grad | e 🖟 | | |
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | • | RENAL/GENITO | DURINARY | | |
| Bladder späsms | absent | mild symptoms,<br>not requiring<br>intervention | symptoms<br>requiring<br>antispasmotic | severe symptoms<br>requiring<br>narcotic | - |
| Creatinine | WNL | > ULN - 1.5 x<br>ULN | > 1.5 - 3.0 x ULN | > 3.0 - 6.0 x ULN | > 6.0 x ULN |
| Note: Adjust to age-appr | | pediatric patients. | | | |
| Dysuria<br>(painful urination) | none | mild symptoms requiring no intervention | symptoms<br>relieved with<br>therapy | symptoms not<br>relieved despite<br>therapy | - |
| Fistula or GU fistula<br>(e.g., vaginal,<br>vesicovaginal) | none | - | - | requiring<br>intervention | requiring<br>surgery |
| Hemoglobinuria | - | present | - | - | 48 |
| Hematuria (in the abse | ence of vaginal b | | | category. | |
| Incontinence | none | with coughing, sneezing, etc. | spontaneous,<br>some control | no control (in the absence of fistula) | • |
| Operative injury to bladder and/or ureter Proteinuria Note: If there is an incorrect Renal failure Ureteral obstruction | none normal or < 0.15 g/24 hours onsistency betweenone none | 1+ or 0.15 - 1.0<br>g/24 hours<br>een absolute value and<br>-<br>unilateral, not<br>requiring surgery | injury of bladder with primary repair 2+ to 3+ or 1.0 - 3.5 g/24 hours d uristix reading, use | sepsis, fistula, or obstruction requiring secondary surgery; loss of one kidney; injury requiring anastomosis or re-implantation 4+ or > 3.5 g/24 hours | septic obstruction of both kidneys or vesicovagin al fistula requiring diversion nephrotic syndrome or grading. requiring dialysis and irreversible stent, nephrostom y tube, or |
| Urinary electrolyte wasting (e.g., Fanconi's syndrome, renal tubular acidosis) Also consider Acidosis Urinary frequency/urgency | none<br>s, Bicarbonate, H<br>normal | asymptomatic, not requiring treatment [ypocalcemia, Hypop] increase in frequency or nocturia up to 2 x normal | mild, reversible and manageable with oral replacement hosphatemia. increase > 2 x normal but < hourly | reversible but requiring IV replacement hourly or more with urgency, or requiring catheter | surgery irreversible, requiring continued replacement |

| | | Grade | | rage | |
|---|---|---|---|---|---|
| | | Grade | е . | | |
| Toxicity Urinary retention | 0<br>normal | hesitancy or | 2<br>hesitancy | requiring | 4<br>bladder |
| | | dribbling, but no significant residual urine; retention occurring during the immediate postoperative period | requiring medication or occasional in/out catheterization (<4 x per week), or operative bladder atony requiring indwelling catheter beyond immediate postoperative period but for < 6 weeks | frequent in/out catheterization (≥ 4 x per week) or urological intervention (e.g., TURP, suprapubic tube, urethrotomy) | rupture |
| Urine color change (not related to other | normal | asymptomatic,<br>change in urine | - | - | • |
| dietary or physiologic cause e.g., bilirubin, concentrated urine, hematuria) | | color | | | |
| Vaginal bleeding is gra | aded in the HEMO | | | | |
| Vaginitis<br>(not due to infection) | none | mild, not<br>requiring<br>treatment | moderate,<br>relieved with<br>treatment | severe, not<br>relieved with<br>treatment, or<br>ulceration not<br>requiring surgery | ulceration<br>requiring<br>surgery |
| Renal/Genitourinar<br>y-Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| <del></del> | | SECONDARY MA | LIGNANCY | | |
| Secondary Malignancy-Other (Specify type,) excludes metastastic tumors | none | _ | _ | _ | present |
| | SF | XUAL/REPRODUC | TIVE FUNCTION | | |
| Dyspareunia is gradeo<br>Dysmenorrhea is grad | l in the PAIN cate | gory. | | | |
| Erectile impotence | normal | mild (erections | moderate | no erections | _ |
| - | | impaired but<br>satisfactory) | (erections impaired, unsatisfactory for intercourse) | | |
| Female sterility | normal | - | _ | sterile | - |
| Femininization of male | | | | | |
| Irregular menses<br>(change from<br>baseline) | normal | occasionally irregular or lengthened interval, but continuing menstrual cycles | very irregular,<br>but continuing<br>menstrual cycles | persistent<br>amenorrhea | |

| | | Grad | le 💀 | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Libido | normal | decrease in interest | severe loss of interest | - | • |
| Male infertility | - | · · <u>-</u> | Oligospermia<br>(low sperm<br>count) | Azoospermia<br>(no sperm) | - |
| Masculinization of fen | nale is graded in | the ENDOCRINE ca | tegory. | | |
| Vaginal dryness | normal | mild | requiring<br>treatment and/or<br>interfering with<br>sexual function,<br>dyspareunia | - | - |
| Sexual/Reproductiv e Function-Other (Specify,) | none | mild | moderate | severe | disabling |
| | SYND | ROMES (not include | d in previous catego | ries) | |
| Acute vascular leak sy | | | | | |
| ARDS (Adult Respirat | tory Distress Syr | ndrome) is graded in t | the PULMONARY ca | tegory. | |
| Autoimmune reaction | s are graded in t | he ALLERGY/IMMU | JNOLOGY category. | | |
| DIC (disseminated int | ravascular coag | ulation) is graded in t | he COAGULATION | category. | |
| Fanconi's syndrome is | graded as Urin | ary electrolyte wastin | g in the RENAL/GE | NITOURINARY cate | gory. |
| Renal tubular acidosis | ie graded as Ur | inary electrolyte wast | ing in the RENAL/C | ENITOURINARY | etegory |
| Stevens-Johnson synd | rome (exithems | multiforma) is arada | d in the DERMATOL | OCV /SKINI catogor | r chory. |
| Sievens-Johnson synd | tome (erymema | (idiametrale programa) | u mine Denvia | OCDINE antonomy | у. |
| SIADH (syndrome of | inappropriate ar | maiurenc normone) | is graded in the END | OCKINE category. | |
| Thrombotic microangs<br>syndrom/HUS) is gra | opathy (e.g., thi<br>ded in the COA | GULATION category | • | | |
| Tumor flare | none | mild pain not interfering with function | moderate pain; pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain; pain or analgesics interfering with function and interfering with activities of daily living | Disabling |
| therapy (e.g., ant inflammation of | s characterized b<br>i-estrogens/and<br>visible tumor, h | y a constellation of sy<br>rogens or additional<br>ypercalcemia, diffuse | hormones). The symp | otoms/signs include<br>electrolyte disturba | tumor pain, |
| Tumor lysis<br>syndrome | absent | - | - | present | - |
| Also consider Hyperk<br>Urinary electrolyte wa<br>RENAL/GENITOURI | sting (e.g., Fanc | oni's syndrome, rena | l tubular acidosis) is { | graded under the | - |
| Syndromes-Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |

## Toxicity Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| Toxicity: | Date of Treatment: | | Course Number: | |
|---|---|---|---|---|
| Date of onset: | 0 | | Grade at onset: | |
| Date of first change in grade: | | | Grade: | |
| Date of next change in grade: | | | Grade: | |
| Date of next change in grade: | | | Grade: | |
| Date of next change in grade: | | | Grade: | |
| Date of next change in grade: | | | Grade: | |
| Date of next change in grade: | | | Grade: | |
| Did toxicity resolve? | Yes | No | | |
| If so, date of resolution of toxicity: | | | | |
| Date of last observation (if prior to | | | | |
| recovery): | | | | |
| Reason(s) observations stopped (if | | | | |
| prior to recovery): | | | | |
| Was patient retreated? | Yes | No | | |
| If yes, was treatment delayed for | | | | |
| recovery? | Yes | No | | |
| Date of next treatment? | | | | |
| Dose reduced for next treatment? | Yes | No | | |
| Additional Comments: | ¥ | | | |
| If module is being activated for new to grading: Grade 0 = | | | | ity |

## Infection Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent. 1. Use the Common Toxicity Criteria definitions to grade the severity of the infection. 2. Specify type of infection from the following (CHŎOSE ONE): BACTERIAL **FUNGAL PROTOZOAL** VIRAL UNKNOWN 3. Specify site of infection from the following (CHOOSE ALL THAT APPLY): **BLOOD CULTURE POSITIVE BONE INFECTION** CATHETER (intravenous) CATHETER (intravenous), tunnel infection CENTRAL NERVOUS SYSTEM INFECTION EAR INFECTION EYE INFECTION **GASTROINTESTINAL INFECTION** ORAL INFECTION **PNEUMONIA** SKIN INFECTION UPPER RESPIRATORY INFECTION URINARY TRACT INFECTION VAGINAL INFECTION INFECTION, not otherwise specified (Specify site, \_\_\_\_\_) 4. Specify organism, if known: 5. Prophylactic antibiotic, antifungal, or antiviral therapy administration \_\_\_\_No\_ If prophylaxis was given prior to infection, please specify below: Antibiotic prophylaxis \_\_\_\_\_ Antifungal prophylaxis

Antiviral prophylaxis

Other prophylaxis
#### APPENDIX E

# DISPENSING AND OTHER INFORMATION FOR IDEC-C2B8 (Rituximab)

**DESCRIPTION:** IDEC-C2B8 is a mouse/human chimeric antibody. The IDEC-C2B8 antibody is produced by a Chinese hamster ovary transfectoma.

#### RECOMMENDED PREPARATION AND ADMINISTRATION:

- 1) Refer to the clinical trial protocol for details about the dose and dose schedule.
- 2) Storage:
  IDEC-C2B8 should be stored at 2-8 °C. Do not freeze or store at room temperature. The products is a protein -- HANDLE GENTLY AND AVOID FOAMING. The avoidance of foaming during product handling, preparation and administration is important, as foaming may lead to the de-naturing of the product proteins.
- 3) All transfer procedures require strict adherence to aseptic techniques, preferably in a laminar flow hood.
- 4) Reconstitution and Dilution of IDEC-C2B8 (rituximab):
  - a. Refrigerate (2-8 °C) all materials and solutions prior to use.
  - b. Use sterile, non-pyrogenic, disposable containers, syringes, needles, stopcocks and transfer tubing, etc.
  - c. Using a sterile syringe and a 21 gauge or larger needle, transfer the necessary amount of rituximab from the vial into a partially filled IV pack containing sterile, pyrongen free 0.9% Sodium Chloride, USP (saline solution). The final concentration of rituximab should be approximately 1 mg/mL. Mix by inverting the bag gently.

For lots 0122-0125 the final preparation should be administered through a 0.22 micron low-protein binding in line filter, such as IMED 9216, into the outflow port of the bag containing the infusion solution. For other lots this will not be required.

Caution should be taken during the preparation of the drug. (see Appendix I). Parental drug products should be inspected visually for particulate matter prior to administration, Preparations of rituximab containing visible particles should note be used. As with all parenteral drug products, aseptic procedures should be used during the preparation and administration of rituximab.

NOTE: DO NOT USE A VACUUM APPARATUS to transfer IDEC-C2B8 from the syringe to the infusion pack. DO NOT USE evacuated glass container which require vented administration sets, because this causes foaming when air bubbles pass through the solution.

5) The administration of IDEC-C2B8 will be accomplished by slow IV infusion. CAUTION: DO NOT ADMINISTER AS AN INTRAVENOUS PUSH OR BOLUS.

- 6) IV pumps such as the IMED 960 may be used with the IDEC-C2B8 infusion. DO NOT INFUSE CONCURRENTLY with another IV solution or IV medications. Prime the line with the IDEC-C2B8 solution such that approximately 30 mL are delivered. This will saturate the filter and tubing.
- 7) If a delay in administration of the infusion occurs after the product is prepared, the properly identified container may be kept refrigerated at 2-8 °C for up to six hours.

#### **OCCUPATIONAL SAFETY**

Study medication are not expected to pose significant occupational safety risks to investigational staff under normal conditions of use and administration. However, precautions should be taken to avoid direct contact with study medication.

#### **ADVERSE CLINICAL EVENTS:**

Throughout the course of the study, every effort should be made to remain alert to possible adverse experiences. Adverse events should be recorded using the toxicity criteria as stated in Appendix D. In the event of an adverse experience, appropriate medical intervention should be provided and necessary, the investigational agent (IDEC-C2B8 [rituximab]) should be discontinued.

1) Infusion Related Adverse Events
An infusion-related symptom complex consisting primarily of fever and chills/rigors can occur predominantly during the first IDEC-C2B8 infusion, usually within the first two hours. Other infusion-related symptoms include nausea, urticaria/rash, fatigue, headache, pruritus, sensation of tongue or throat swelling, rhinitis, vomiting, flushing, and pain at disease site. The incidence of infusion-related events decreases dramatically with subsequent infusions.

Transient hypotention and bronchospasm have occurred in association with IDEC-C2B8 infusion as a component of an infusion-related symptom complex. Patients with preexisting pulmonary disease may have an increased risk of bronchospasm. These symptoms are usually reversible with temporary interruption of the IDEC-C2B8 infusion and administration of acetaminophen, diphenhydramine intravenous saline or bronchodilators. The infusion may be completed when symptoms abate.

Patients with a history of cardiac disease (i.e., angina, cardiac arrhythmias, or congestive heart failure) should be monitored closely.

Anaphylactoid and other hypersensitivity reactions can occur following the IV administration of proteins to patients. Medications for the treatment of hypersensitivity reactions, e.g., epinephrine, antihistamines, should be available for immediate use in the event of an allergic reaction during administration.

2) Hematologic

Following are the results of an integrated safety analysis with 282 patients treated with single agent IDEC-C2B8 at 375 mg/m2.

¥ Neutropenia

During treatment, AGC nadirs were 1000 - 1500/mm3 in 9.2% of patients, 500 - 999/mm3 in 1.4% of patients, and <500 mm3 in 1.1% of patients. During a one year follow-up period, nadirs were 1000 - 1500/mm3 in 6.7% of patients, 500 - 999/mm3 in 5.0% of patients, and <500 mm3 in 2.5% of patients.

¥ Thrombocytopenia

During treatment, platelet values were 50,000-75,000/mm3 in 2.8% of patients and <50,000 in 1.1% of patients. During a one year follow-up period, platelet values were 50,000 - 75,000/mm3 in 1.8% of patients and <50,000 in 0.4% of patients. Two patients received platelet transfusions.

#### ¥ Anemia

During treatment, hemoglobin values were 8-10 gm/dL in 7.8% of patients <8 gm/dL in 2.8% of patients. During a one year follow-up period, hemoglobin values were 8-10 gm/dL in 3.2% of patients and <8 gm/dL in 0.7% of patients. Only four patients required transfusions and two received erythropoietin for anemia. Pure red cell aplasia was reported in one patient.

### 3) Infection

Although IDEC-C2B8 induces B-cell depletion and can be associated with decrease serum immunoglobulins, the incidence of infection does not appear to be greater than expected in this patient population and serious infections were considerably less common than report with conventional chemotherapy [1-7]. During treatment and for up to one year following therapy, approximately 17% an 12%, respectively, of patients developed infections which were usually common, nonopportunistic and Grade 1 or 2.

### 4) Other

There are no known drug interaction with IDEC-C2B8. Patients with HAMA/HACA titers may have allergic or hypersensitivity reactions when treated with other diagnostic or therapeutic antibodies. Positive HACA results were reported in <1% of the patients receiving IDEC-C2B8.

IDEC-C2B8 has not been associated with clinically significant hepatic or renal toxicity, through mild, transient increases in liver function tests have occurred.

Bronchiolitis obliterans was reported in one patient.

#### FOR ADDITIONAL INFORMATION CONTACT:

Clinical Trials Management, IDEC Pharmaceuticals Corporation, 11011 Torreyana Road, San Diego, CA 92121. Telephone: (800)447-4131.

# Appendix F

#### Additional Safety Guidelines for Use of Interferon

Consider for exclusion from interferon therapy, or dose modification, according to these guidelines (discuss with P.I.):

#### **Inclusion Criteria**

Patients should be assessed for adequate organ function as follows:

Hematologic: WBC  $\geq$  3,000/mm<sup>2</sup> (Neutrophils  $\geq$  15

WBC  $\geq$  3,000/mm<sup>2</sup> (Neutrophils  $\geq$  1500/mm<sup>3</sup>); platelets  $\geq$  70,000/mm<sup>3</sup>; Hemoglobin 10.0

gm% or 8.21 mmol/L. For hematologic malignancies these inclusion criteria are at the

discretion of the investigator

Hepatic: Bilirubin < 2.0 mg% cr 34.2 umol/L; SGOT or SGPT < 3.0 X's upper limit of normal;

alkaline phosphatase < 3.0 X's upper limit of normal. Patients whose SGOT, SGPT or

alkaline phosphatase are elevated as a result of metastatic disease are eligible.

Renal Serum creatinine: within normal limits.

There should be no acute infection requiring systemic antibiotics.

Patients with diabetes or hypertension should be considered for a baseline ocular examination.

#### **Exclusion Criteria**

- 1) Patients with a history of hypersensitivity to interfeorn alfa or any component of the injection.
- Patient with pre-existing psychiatric condition, especially depression or a history of severe psychiatric disorder.
- 3) Patients with a history of severely debilitating cardiovascular disease, such as unstable angina or uncontrolled congestive heart failure.
- 4) History of severely debilitating pulmonary disease, such as chronic obstructive pulmonary disease.
- 5) Patients with history of diabetes mellitus prone to ketoacidosis.
- 6) Patients with coagulation disorders, such as thrombophlebitis or pulmonary embolism.
- Patients with severe myelosuppression.
- 8) Patients with decompensated liver disease, autoimmune hepatitis or history of autoimmune disease.
- Patients with pre-existing thyroid abnormalities, whose thyroid function cannot be maintained in the normal range.
- 10) Patients with clinically significant retinal abnormalities.

# Appendix G

Guidelines for Filing Reports of Adverse Experience at MDACC

The administration of agents for which MDACC holds the IND confers increased requirements for reporting Adverse Experiences. The responsibility for reporting an AE to the FDA rests with the sponsor of the IND. As holder of the IND, MDACC becomes responsible for the reporting of all Adverse Experiences. It is the responsibility of the individual clinical investigator to report these to the Office of Protocol Research, who in turn is responsible for reporting to the FDA.

#### 1.0 Types of Adverse Experiences

Two types of Adverse Experience requiring reporting to the IRB and IND sponsor are recognized:

- 1. Serious Adverse Experiences
- 2. Unexpected Adverse Experiences

The FDA definitions of these two types are included in Addendum A.

#### 2.0 Serious Adverse Experience

For the majority of trials performed at MDACC, a serious adverse experience is a clinical event occurring subsequent to the administration of an agent or intervention classified as an Investigational New Drug (IND) which can be characterized as fatal, life-threatening, permanently disabling, requiring hospitalization, or an overdose.

It is recognized that in many instances it may not be possible to absolutely determine whether a clinical event is due to the IND or to progressive cancer. In these instances, a report should be filed, indicating the unlikelihood of a causal relationship.

#### 2.1. Fatal Reactions

Although no specific time period is specifically defined in the regulations, historically, an AE report has been required if a patient expires within 30 days of receiving an investigational new drug or treatment. Although the clinical scenario may suggest an early death secondary to rapidly progressing disease, this event should be reported since the possibility of the agent contributing to this adverse event cannot be excluded.

#### 2.2 Life-threatening

By definition, any grade 4 toxicity using the Common Toxicity Scale is life-threatening and should be reported when they occur in a patient receiving an investigational new drug. A grade 3 reaction, associated with significant co-morbid conditions, might also be life-threatening and should be reported, e.g. grade 3 vomiting leading to renal failure in a patient with compromised kidneys.

#### 2.3 Permanently Disabling

If an IND agent is administered in a situation where prolonged survival is possible, and permanent damage or sequelae occurred sufficient to significantly compromise normal function an adverse experience report should be filed. Example might include marrow aplasia resulting in transfusion-dependency, or pulmonary fibrosis leading to symptomatic restrictive pulmonary disease.

#### 2.4 Hospitalization

Although no time period is specified in the regulations, hospitalization or prolongation of hospital stay within 30 days or receiving an IND agent or intervention must be reported. If the hospitalization is incidental to an event unrelated to the drug administration or the underlying disease, e.g. fracture secondary to a fall, an AE report should still be filed.

#### 2.5 Overdose

Any dose greater than 25% above the protocol specified dose should be reported with a description of the resultant side-effects or toxicity.

#### 3.0 Unexpected Adverse Experience

An unexpected adverse experience is a clinical event that is not identified in nature, severity, or frequency in the investigator's brochure, protocol, or other pertinent supporting literature. At times, the occurrence of an unexpected adverse experience might not be suspected until more than one event has occurred, e.g. multiple cases of herpes zoster in a small phase II trial. Once the clinical event has been identified, all cases should be reported. No degree of unexpected toxicity is specified, but practically, it is unusual to be able to discern < grade 2 toxicity.

- 4.0 Schedule of Required Reports of Adverse Experiences
- A. Serious and/or Unexpected AE

Submit a written report to the Office of Protocol Research within 10 working days of the adverse experience.

Unexpected fatal or life-threatening experiences must be phoned immediately to the Office of Protocol research at ext. 2-2933. OPR will notify the FDA within 3 working days. A follow-up written report should be submitted to OPR within 10 working days.

B.- Not serious and/or not Unexpected AE For MDACC sponsored INDs only

Submit written reports to OPR every month. OPR will submit this information in the annual IND report submitted to the FDA.

#### Addendum A

#### A. Serious Adverse Experience

"Any experience that suggests a significant hazard, contradiction, side effect or precaution, including any experience that is fatal, life-threatening, is permanently disabling, requires inpatient hospitalization or is a congenital anomaly, cancer or overdose. This definition also encompasses results obtained from tests in lab animals suggesting a significant risk for human subjects, including any finding mutagenicity, teratogenicity or carcinogenicity".

#### B. Unexpected Adverse Experience

"Any adverse experience that is not identified in nature, severity or frequency in the current investigator brochure or if an investigator's brochure is not required, that is not identified innature, severity or frequency in the risk information described in the general investigational plan or elsewhere in the current application".

#### Addendum B

A. Reporting requirements: Genentech requires certain events to be reported to Genentech (MedWatch 3500 form), attached.

#### APPENDIX H

For use by user-facilities, distributors and manufacturers for MANDATORY reporting

| Form Approved | See OMB statement on revers |
|------------------|-----------------------------|
| Mir report # | a mentant ou lavers |
| UF/Dist report # | |
| - | |

Therapy dates ( if unknown, give duration) irom/to or best estimate

Event abated after use stopped or dose reduced

✓ Yes □ no □ doesn't apply

#1 yes no doesn't

≥ yes no doesn't

2. Phone number

3. Report Source (check all that apply) kreign ☐ study ☐ iterature Consumer

user facility

Company representative

distibutor cther:

☐ yes

□ you

Event responsed after reintroduction

#1:

**#2**:

Page 💆 Patient Information C. Suspect medication(s) 2. Age at time of event: 4. Weight 1. Harne (give labeled strength & mir/scheler, if kno [ ferrale **#1**or male [ **\$2** kg 2. Doss, frequency & route used B. Adverse event or product problem 1. Adverse Event and/or Product Problem (e.g. defects/malfunctions) 2. Outcomes attributed to adverse event 42: (check all that apply) ☐ deability 4. Diagnosis for use (Indication) death:\_\_ congential anomaly #1; ☐ life-threatening required intervention to prevent permanentimperment/damage 6. Late (d known) hospitalization - mitial or prolonged 7. Exp date (# known) C other: #1: #1: #2 **\$2** . 3. Date of 4. Date of this report (mo/day/yr) (morday/yri 9. NDC# - for product problems only (if known) 5. Describe event or problem 10. Concomitant medical products and therapy dates (exclude treatment of event) G. All manufacturers 1. Contact office - name/address (& miring site for devices) Date received by manufacturer morday/yr A(NOA) #\_ ND# 8. Relevant tests/isboratory data, including dates 5. If IND, protocol # PLA#\_ pre-1938 7. Type of report (check all that apply) OTC product ☐ 5-day ☐ 15-day 8. Adverse event term(s) ☐ 10-day ☐ periodic Initial I follow-upst Other relevant history, including preexisting conditions (e.g., allergies, race, pregnancy, smoking and alcohol use, hepatichensi dysfunction, etc.) 9. Mfr. report number E. Initial Reporter 1) Name, address & phone #



Submission of a report does not constitute an admission that medical personnel, user facility, distributor, manufacturer or product caused or contributed to the event.

| 2. Health professional? | 3. Occupation | 4. Initial reporter aiso sent report to FDA | | |
|---|---|---|---|---|
| | | ☐ yes | □ m | unk |
| DEC Safety Review Of | ficer: | | | |

2. Health professional?

# The University of Texas M.D. ANDERSON CANCER CENTER

INFORMED CONSENT FOR PARTICIPATION IN RESEARCH

PROTOCOL TITLE: FLUDARABINE, MITOXANTRONE, AND

**DEXAMETHASONE (FND) PLUS ANTI-CD20** 

**MONOCLONAL ANTIBODY (IDEC-C2B8) FOR STAGE** 

IV INDOLENT LYMPHOMA

| 4 | |
|--------------------|-------------|
| Participant's Name | I.D. Number |

You are being asked to take part in this clinical research study at The University of Texas M.D. Anderson Cancer Center (hereinafter referred to as "UTMDACC"). Clinical studies include only individuals who choose to take part. This consent form explains why we are performing this research study and what your role would be should you choose to participate. This form also describes the possible risks linked with being in this study. After reviewing this information with the registering personnel, you should know enough about this study to be able to make an informed decision on whether you want to be in the study. This study complies with all laws and regulations that apply.

You are being asked to take part in this study because you have Stage IV indolent lymphoma.

# **DESCRIPTION OF RESEARCH**

- 2. PURPOSE OF STUDY: The goal of this clinical research study is to compare chemotherapy given with rituximab to chemotherapy followed by rituximab. The safety of both treatment schedules will be studied. Laboratory tests of genetic changes in blood and bone marrow before and during the study will also be monitored.
- 3. **DESCRIPTION OF RESEARCH:** Rituximab seeks out and helps destroy cancer cells.

Before treatment starts, patients will have a complete exam, including blood and urine tests. Chest x-rays and CT scans will be done. Bone marrow samples will be taken; this is done with a large needle. Tests of heart function and lung function will be done. Tumors and lesions will be measured.

Patients in this study will be assigned at random (as in the toss of a coin) to 1 of 2 groups. Each group will receive 8 cycles of treatment. One cycle will last 28 days.

Most of the drugs are given by vein. A catheter (a tube) will be placed in a vein to decrease the number of needle sticks. Dexamethasone may be taken by mouth instead of given by vein.

Patients in group 1 will receive the drug rituximab on Days 1 and 8 of the first course, and on Day 1 only of Cycles 2-5 of FND. Fludarabine will be given on Days 2-4, mitoxantrone on Day 2, and dexamethasone on Days 1-5 of each 28-day cycle (FND). Patients in group 1 will not receive rituximab in Cycles 6 - 8. When the 8 cycles are finished, patients will begin receiving the drug interferon on Days 1-14 each month for 1 year. Dexamethasone will be given on Days 1-3 every month for 1 year.

Patients in group 2 will receive fludarabine on Days 1-3, mitoxantrone on Day 1, and dexamethasone on Days 1-5 of each 28-day cycle. When 8 cycles of treatment are finished, patients will begin receiving the drug interferon on Days 1-14 each month for 1 year. Dexamethasone will be given on Days 1-3 every month for 1 year. About 4 months after interferon treatment starts, patients in group 2 will begin receiving rituximab once a month for 6 months.

Other drugs may be given to help decrease the risk of or ease side effects. Treatment may be delayed or stopped if side effects are severe.

Some patients in this study, with changes in certain genes will receive different chemotherapy drugs than other patients in the study will. The patients will, like all the other patients, receive rituximab and interferon. But instead of the FND chemotherapy regimen, they will receive a sequence of three regimens, CHOD-Bleo, ESHAP, and NOPP. The drugs in these regimens include: cyclophosphamide, doxorubicin, vincristine, bleomycin, VP-16, Ara-C, cisplatin, mitoxantrone, procarbazine, and corticosteroids (prednisone, methylprednisolone, dexamethasone).

During the study, patients will have blood tests every week. Complete exams will be given in Cycles 2 and 4; patients will return to the clinic for these. Every 2 or 3 cycles, patients will have a chest x-ray and CT scans of the abdomen and pelvis. Bone marrow samples will be taken. Heart function tests (EKG) will be done as needed.

After the study ends, patients will return for checkups every 3 months in the first year, every 4 months in years 2 and 3, and every 6 months in years 4 and 5. After that, checkups will be needed once a year. Blood and bone marrow samples will be taken at these visits.

This is an investigational study. Rituximab is approved by FDA for commercial use. The other drugs used in the study are also approved for commercial use. About 210 patients will take part in the study. All will be enrolled at UTMDACC. Genentech, Inc., the makers of rituximab, will work with patients or their insurance companies to insure that no one is excluded from the study for money reasons. The protocol is partially funded by research grants from Genentech, Inc., Integrated Therapeutics Group, Inc., and Immunex Corporation.



4. RISKS, SIDE EFFECTS AND DISCOMFORTS TO PARTICIPANTS: Fludarabine, mitoxantrone, dexamethasone, and interferon may cause low blood cell counts (white blood cells, red blood cells, and platelets). This means that while participants take the drugs, there is more of a chance of getting an infection, including pneumonia. Participants may become anemic and/or have problems with bleeding, bruising, fatigue, and/or shortness of breath. Participants may need a blood transfusion. Participants may die. These drugs may cause upset stomach, nausea, vomiting, diarrhea, mouth ulcers, and/or hair loss. The drugs may cause heart damage. The patient may have a fever, bone pain, and/or fluid retention, causing swelling.

Rituximab may cause fever, chills, nausea, and vomiting. The patient may have a rash, headache, muscle aches, and/or swelling from fluid buildup. The patient may feel dizzy and/or tired. Hives, breathing trouble, low blood pressure, and/or sweating may occur. There may be tenderness and/or swelling at tumor or lesions sites. Allergic reactions, including low blood pressure, shortness of breath, and/or wheezing, which can be fatal, may occur. These severe reactions have occurred with the first dose of rituximab, so this dose (especially) is monitored carefully and given slowly. Severe skin rashes, which can be fatal, may occur.

Rituximab does temporarily decrease one normal blood cell element (B-cells), and this can result in some decreased resistance to certain types of infections, such as viruses. There is also a temporary decrease of immunoglobulin levels, which can also lower the resistance of the body to infections.

Using these drugs together may cause other side effects that are not seen when each drug is given alone.

Participants may experience pain, bleeding, and/or bruising from the blood draws or bone marrow tests. Participants may faint and/or develop an infection with inflammation of the vein at the site where blood is drawn.

This clinical research study may involve unpredictable risks to the participant.

- 4a. Participants must practice birth control during the study if they are sexually active. There could be unknown risks to an unborn child or the patient. If the patient is pregnant, she may not participate in this study. Mothers should refrain from breast-feeding during the study to avoid injury to their children.
- 5. **POTENTIAL BENEFITS:** Treatment on this study may shrink or slow the growth of the tumor. There may be no benefits at all for patients in the study. Future patients may benefit from what is learned.
- 6. ALTERNATE PROCEDURES OR TREATMENTS: Individuals may choose not to take part in this study. Individuals may choose to be treated with a standard chemotherapy drug such as chlorambucil or combinations such as CVP or CHOP. If the tumors are not large or threatening, individuals may choose only to be observed by their doctors. Individuals may choose to receive other investigational therapy, if available. Individuals



can choose not to have treatment for cancer at all. In all cases, individuals will receive care for symptoms and pain.

# I understand that the following statements about this study are true:

- 7. According to the M.D. Anderson Cancer Center conflict of interest policy, the principal investigator of this study and the participant's primary physician cannot have a financial interest in any aspect of this research. However, because of the unconditional priority of patient care, a circumstance may arise wherein a participant may need to be cared for by a physician and/or administrator who does have some form of financial interest in the sponsor of this study.
- 8. If at any time I wish to acquire further updated information regarding the financial interests of any physician and/or administrator here who has cared for me, I may call the Office of Research Administration at (713) 745-1697. Upon request, I will be given access to information disclosing the identity of all physicians and/or administrators who have a financial interest in the sponsor of this study.
- 9. My participation is voluntary.
- 10. I may ask any questions I have about this study, including financial considerations, of my physician Dr. \_\_\_\_\_\_. I may also contact the principal investigator for this study Dr. Peter McLaughlin at (713) 792-2860 or the Chairman of UTMDACC's Surveillance Committee at (713) 792-2933 with any questions that have to do with my rights.
- 11. I may withdraw at any time without any penalty or loss of benefits. I should first discuss leaving the study with my physician. Should I withdraw from this study, I may still be treated at UTMDACC by my physician.
- 12. This study may be changed or stopped at any time by my doctor, the principal investigator, the study sponsor, or the Surveillance Committee of UTMDACC.
- 13. I will be informed of any new findings that might affect my willingness to continue participating in the study.
- 14. UTMDACC will take appropriate steps to keep my personal information private. However, there is no guarantee of absolute privacy. The Food and Drug Administration ("FDA"), Genentech, Inc., Integrated Therapeutics Group, Inc., and Immunex Corporation might review my record to collect data or to see that the research is being done safely and correctly.
  - Under very rare circumstances, the FDA could be required to reveal the names of participants.
- 15. If I suffer injury as a result of participation in this study, the institution will provide reasonable medical care. I cannot expect to receive reimbursement of expenses or financial compensation from the institution, the sponsorement

\*IRB Approved Consent

\* Date of Approved 1-29-6

\*Signature Mac Month

Protocol DM97-261 Revised January 8, 2002 Page 5 of 6

manufacturer for this injury. I may also contact the Chairman of UTMDACC's Surveillance Committee at 713-792-2933 with questions about study related injuries.

- 16. Unless I am told otherwise, all of the costs linked with this study are to be paid by me or the 3<sup>rd</sup> party payer (HMO, Health Insurance company, etc.) responsible for my health care expenses. If medications or devices are provided for free or at a reduced cost, I will not be charged or will pay a reduced charge for that item.
- 17. I recognize that there are no plans to provide any compensation to me for any patents or discoveries that may result from my participation in this research.
- 18. All participants must practice birth control. Female participants should not breast feed their infants. If a female participant becomes pregnant, or suspects that she is pregnant, she must notify her physician-immediately. Getting pregnant may result in my removal from participation in this study.

<sup>\*</sup>IRB Approved Consent

<sup>\*</sup> Date of Approved\_

<sup>\*</sup>Signature mance month

# **CONSENT**

| questions about this study and reflect an | and having had the chance to ask all my add consult with any others that I might like to, I to enroll me on this study. I have been given |
|---|---|
| DATE | SIGNATURE OF PARTICIPANT |
| WITNESS OTHER THAN PHYSICIAN OR INVESTIGATOR | SIGNATURE OF PERSON RESPONSIBLE & RELATIONSHIP |
| authorized representative, using a langu believe that I have fully informed this par | audy with the participant and/or his or her age that is understandable and appropriate. In ticipant of the nature of this study and its the participant understood this explanation. |
| PHYSICIAN/INVESTIGATOR | |
| I have translated the above informed cor<br>participant. | nsent into for this (Name of Language) |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR & DATE |

<sup>\*</sup>Edited
\*IRB Approved Consent
\* Date of Approved /-292
\*Signature Management